

An Open-Label Safety Study of USL261 in the Outpatient Freatment of Subjects with Seizure Clusters

Protocol Number P261-402, and an open-Label Subjects with Seizure Clusters Upsher-Smith Laboratories, Inc.

This document cannot be used to support any mark 6701 Evenstad Drive Maple Grove, MN 55369

**Date of Plan:** 15MAY2017 (v2.0)

**CONFIDENTIAL** 

### STATISTICAL ANALYSIS PLAN

### Final v2.0

An Open-Label Safety Study of USL261 in the Outpatient Treatment of Subjects with Seizure Clusters



## **TABLE OF CONTENTS**

| LIST OF A | BBREVIATIONS | .5 |
|---|---|---|
| 1. | INTRODUCTION | .6 |
| 2. | STUDY DESIGN | .60 |
| 2.1. | General Study Design and Plan | 36 |
| 2.2. | Randomization and Method of Treatment Assignment | 10 |
| 2.3. | Study Procedures | 10 |
| 3. | STUDY OBJECTIVES AND CLINICAL ENDPOINTS | 13 |
| 3.1. | Study Objectives | 13 |
| 3.2. | Clinical Endpoints | 13 |
| 3.2.1. | Safety Endpoints | 13 |
| 3.2.2. | Efficacy Endpoints | 13 |
| 3.2.3. | Exploratory Efficacy Endpoints | 13 |
| 3.2.4. | Outcome Endpoints | 14 |
| 4. | STUDY DESIGN General Study Design and Plan Randomization and Method of Treatment Assignment Study Procedures STUDY OBJECTIVES AND CLINICAL ENDPOINTS Study Objectives Clinical Endpoints Safety Endpoints Exploratory Efficacy Endpoints Outcome Endpoints ANALYSIS POPULATIONS Enrolled Population Safety Population Safety Evaluable Population GENERAL STATISTICAL CONSIDERATIONS | 14 |
| 4.1. | Enrolled Population | 14 |
| 4.2. | Safety Population | 14 |
| 4.3. | Efficacy Evaluable Population | 14 |
| 5. | | |
| 5.1. | General Consideration | |
| 5.2. | Baseline | 14 |
| 5.3. | Handling of Missing Data | 15 |
| 5.4. | Interim Analysis | |
| 5.5. | Data and Safety Monitoring Board (DSMB) | 16 |
| 5.6. | Multiple Comparisons and Multiplicity | 16 |
| 5.6.<br>6. 6.1. 10 <sup>0</sup><br>6.1. 10 <sup>0</sup><br>6.2. | STATISTICAL ANALYSIS | 16 |
| 6.100 | Subject Disposition | 16 |
| 6.2. | Treatment Exposure and Treated Seizure Clusters | 16 |
| 6.3. | Protocol Deviations | 17 |
| 6.4. | Demographics and Baseline Characteristics | 17 |
| 6.5. | Medical and Surgical History | 18 |
| 6.6. | Prior and Concomitant Medications | 18 |

| 6.7. | Analyses of Efficacy and Outcome Endpoints | 19 |
|---|---|---|
| 6.7.1. | Efficacy Endpoint | 19 |
| 6.7.2. | Exploratory Efficacy Endpoints | 21 |
| 6.7.3. | Subject and Caregiver Outcome Assessments | 23 |
| 6.8. | Safety Analyses | 24 |
| 6.8.1. | Subject and Caregiver Outcome Assessments Safety Analyses Adverse Events (AEs) | 25 |
| 6.8.2. | Requirement for Unscheduled ER or EMS Visit | 27 |
| 6.8.3. | Columbia-Suicide Severity Rating Scale (C-SSRS) | 27 |
| 6.8.4. | Requirement for Unscheduled ER or EMS Visit | 28 |
| 6.8.5. | Olfactory testing with Brief Smell Identification Test (B-SIT) | 28 |
| 6.8.6. | Laboratory Parameters | 28 |
| 6.8.7. | Vital Signs / Weight | 29 |
| 6.8.8. | Caregiver-Recorded Respiration Rate | 29 |
| 7. | DEVIATIONS FROM THE PROTOCOL SPECIFIED ANALYSIS | 29 |
| 8. | MOCK TABLES, FIGURES, AND DATA LISTINGS | 29 |
| 9. | REFERENCES | 30 |
| Appe | MOCK TABLES, FIGURES, AND DATA LISTINGS REFERENCES ndix 1 Potentially Clinically Significant Laboratory Values | 31 |
| Appe | ndix 2List of AEs of special interest | 32 |
| This document cann | ndix 2 List of AEs of special interest | |

## LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|---|---|
| μL | Microliter |
| AE | Adverse event |
| AED | Antiepileptic Drugs |
| ATC | Anatomia Therenoutic Chemical |
| B-SIT | Brief Smell Identification Test |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| CI | Confidence interval |
| CRO | Contract Research Organization |
| DSMB | Data and Safety Monitoring Board |
| EMS | Brief Smell Identification Test Columbia-Suicide Severity Rating Scale Confidence interval Contract Research Organization Data and Safety Monitoring Board Emergency Medical Services Emergency Room Early Termination Intranasal Interactive Response Technology |
| ER | Emergency Room |
| ET | Early Termination |
| IN | Intranasal |
| IRT | Interactive Response Technology |
| ITI | Intranasal Therapeutics, Inc. |
| ITIQ | Intranasal Therapy Impact Questionnaire |
| IV | Intravenous |
| LAR | Legally acceptable representative |
| MCS | Mental Health Component Score (SF-12v2) |
| Mg | Milligram |
| MedDRA | Medical Dictionary for Regulatory Activities |
| PCI | Potentially clinically important |
| PCS | Potentially clinically significant |
| PHCS | Physical Health Component Score (SF-12v2) |
| PK | Pharmacokinetic |
| PMP PT SF-12v2 SAS SD USL USL 26k | Patient Management Plan |
| PT | Preferred Term in MedDRA |
| SF-12v2 | SF-12v2 Health Survey |
| SAS | Statistical Analysis Software |
| SD S | Standard deviation |
| USL 💉 | Upsher-Smith Laboratories, Inc. |
| USL2012 | intranasar inidazoram, study drug (formerry 111 111) |
| SOC | System Organ Class in MedDRA |
| TEXE | Treatment-emergent adverse event |
| TSQM | Treatment Satisfaction Questionnaire for Medication |
| VNS | Vagus Nerve Stimulator |
| WHO | World Health Organization |
| ine. | |
| Cn. | |
| 80 | |
| This document carried WHO | |

#### 1. INTRODUCTION

Acute repetitive seizures and seizure clusters occur in a subset of epilepsy patients. Seizure clusters have distinguishable characteristics that are easily recognized by patients, caregivers, and physicians and include a consistent onset (auras, prodrome) that may be indicative of convulsive or non-convulsive symptoms. Although patients typically recover between seizures, these seizure can last anywhere from minutes to hours. When a cluster of seizures occurs outside a hospital, the patient must often be transported to an acute care facility so medical personnel can administer intravenous (IV) therapy to stop the seizure(s).<sup>2</sup>

The primary goals of seizure cluster treatment are seizure cessation and prevention of seizure recurrence. Acute benzodiazepine treatment is effective for seizure control and often results in rapid seizure cluster termination; however, most treatment options rely on intervention by emergency medical personnel and therefore delay treatment while the patient is transported to a medical facility.<sup>3</sup> The development of an easily administered outpatient treatment of seizure clusters may reduce the need for emergency medical intervention and decrease seizure cluster duration.

This statistical analysis plan covers the detailed procedures for performing statistical analyses and producing tables, listings, and figures in the Phase III study described in Upsher-Smith Laboratories, Inc. Protocol P261-402 (Fifth Issue, Amendment 4, 20 May 2015).

### 2.

# STUDY DESIGN General Study Design and Plan 2.1.

This is an open-label, multicenter, safety extension study of USL261 in subjects with seizure clusters who have completed study P261-401. However if study P261-401 is terminated, subjects who have completed the Test Dose Visit (Visit 2) of study P261-401 will also be eligible to enter this study (P261-402). Each seizure cluster episode will be treated with a single dose of 5.0 mg USL261. A second dose of 5.0 mg USL261 may be given if the seizure cluster has not terminated within 10 minutes after initial study drug administration or if another seizure occurs between 10 minutes and 6 hours after administration of study drug. However, the second dose will not be administered if the subject has a respiratory rate < 8 breaths per minute, requires emergency rescue treatment with assisted breathing or intubation, or has excessive, uncharacteristic sedation (as defined by the investigator in the Patient Management Plan [PMP]). After each USL261-treated seizure cluster episode, the caregiver will call the study center as soon as possible, but no later than 24 hours after USL261 administration.

After obtaining informed consent and determining that the subject meets the eligibility requirements for this study, the subject/caregiver will be provided with enough study drug to treat one seizure cluster episode (1 treatment kit containing two 5.0 mg doses of USL261) at Visit 1. After one USL261-treated seizure cluster, the subject and caregiver will return to the study center for Visit 2 within 120 hours (5 days) of USL261 administration. At Visit 2, the

subject/caregiver will again be provided with enough study drug to treat 1 seizure cluster episode (1 treatment kit containing two 5.0 mg doses of USL261). After one USL261-treated seizure cluster, the subject and caregiver will return to the study center for Visit 3 within 120 hours (5 days) of USL261 administration. At Visit 3 and all subsequent visits (except for the Final Visit or Early Termination Visit) the subject/caregiver will be provided with enough study drug to treat 2 seizure cluster episodes (2 treatment kits, each containing two 5.0 mg doses of USL261). After Visit 3, subjects and caregivers will return to the study center after every second USL261-treated seizure cluster episode. Each of these visits will occur within 120 hours (5 days) after the last USL261 administration. A minimum of 3 days (72 hours) is required between treatments (1 treatment is defined as the use of one or two 5.0 mg doses of USL261 from one study drug treatment kit to treat a single seizure cluster episode). There is no limitation on the total number of seizure cluster episodes treated during the subject's participation in the study.

The duration of each subject's participation will vary and will be up to approximately 4 years from the date of enrollment (Visit 1). After this period, the study duration may be extended until marketing approval or a time period as approved by the Heath Authority where the study is being conducted. The study will be reviewed on an ongoing basis and immediate discontinuation of the study may occur if: a) safety concerns/issues are noted or have arisen during the conduct of the P261-402 study or other USL261 studies, b) USL261 does not demonstrate efficacy in controlled clinical studies, c) a regulatory authority (regardless of country) requests that clinical studies be interrupted or discontinued, or d) USL discontinues or will discontinue development of USL261.

Before any subject is enrolled in this open label extension study, he/she must have completed study P261-401, or, if Study P261-401 has been terminated, subjects must have completed the Test Dose Visit (Visit 2) of study P261-401. Subjects must meet all other eligibility criteria for this study. Since enrollment is limited to subjects who have participated in study P261-401, a maximum of 240 subjects (the planned number of subjects completing the Comparative Phase in P261-401) are expected to enroll into this extension study.

Figure 1 of study flow chart on next page shows the overall study scheme.



Figure 1 Study Flow Chart

<sup>a</sup> Each study drug treatment kit contains two 5.0 mg doses of USL261

<sup>b</sup> Visits will continue until the Final Visit or Early Termination

### Screening

After subjects and their caregivers have provided informed consent (and, when appropriate, assent), subjects will undergo screening procedures at Visit 1 (which may occur at the same time as of up to 28 days after Visit 4 of the preceding double-blind study P261-401). If Visit 1 of this study (P261-402) is on the same day as Visit 4 of study P261-401, the procedures performed at Visit 4 of study P261-401 that are common to Visit 1 will be used for both studies. If Visit 1 for this study (P261-402) is not on the same day as Visit 4 of P261-401, all necessary procedures will be repeated, except for physical exam, neurological exam, nasal exam, and clinical laboratory testing (hematology, serum chemistry and urinalysis). The time between Visit 4 of study P261-401 and Visit 1 of study P261-402 will be a maximum of 28 days. The time between Visit 4 of study P261-401 and Visit 1 of study P261-402 may be extended in certain cases; however, the extension must be approved by the Sponsor or Contract Research Organization (CRO) designee. If an extension is granted for a given

subject, that subject may have to undergo repeat screening laboratory assessments within 28 days prior to dispensing study drug.

### Treatment Phase

Caregivers will administer the first 5.0 mg dose of USL261 at the time of recognition of a seizure cluster that meets study criteria (according to the subject's PMP). A second dose of USL261 5.0 mg may be administered if (a) the treated seizure cluster has not terminated within 10 minutes after the first dose, or (b) another seizure occurs between 10 minutes and 6 hours after administration of the study drug, AND (in both a and b) the subject does not have a respiratory rate < 8 breaths per minute, does not require emergency rescue treatment with assisted breathing or intubation, and does not have excessive, uncharacteristic sedation (as defined by the investigator in the PMP). The caregiver will monitor the subject for 24 hours after study drug administration to record safety and efficacy assessments. The caregiver will call the study center as soon as possible, but no later than 24 hours, after each USL261-treated seizure cluster episode. If seizure cluster activity persists or recurs following the administration of the second dose, caregivers will initiate the rescue protocol as outlined in the subject's PMP.

For Visits 2 and 3, which occur after each of the first 2 USL261-treated seizure cluster episodes, the subject and caregiver will return to the study center within 120 hours (5 days) of study drug administration.

After Visit 3, if the study drug has successfully treated the subject's seizure cluster episodes, the subject has tolerated the study drug treatment well in the judgment of the investigator, and the subject and caregiver have been compliant with the study procedures including completion of the Subject Workbooks and return of the study drug (used and unused), the subject and caregiver will be instructed to return to the study center after every second seizure cluster episode treated with USL261 until the Final Visit or Early Termination. A minimum of 3 days (72 hours) is required between treatments with study drug.

All study drug containers dispensed, whether used or unused, and Subject Workbooks are to be returned at the next study visit throughout the study. The study center will make monthly telephone calls between visits to caregiver(s) and subject (if subject is able to communicate adequately as determined by the investigator) when visits are more than 1 month apart. If 6 months pass without the subject having a seizure cluster episode, the subject and caregiver will be asked to come to the study center for re-training on study procedures.

The subject or caregiver will immediately report to the investigator (or his/her designee) as soon as possible any significant medical event (including events that are life-threatening or that result in death, hospitalization or prolonged hospitalization, persistent or significant disability, or incapacity of the subject) that occurs to the subject from the time written informed consent is obtained until completion of the final study visit or 7 days after last administration of study drug, whichever is later. The subject or caregiver may also call the study center at any time during the study for help or advice regarding study procedures.

ole 1.

ole 1.

ole 1.

ole 1.

ole 1.

The document control be used to support any materials as provided in a policy of the support of the s

 Table 1
 Schedule of the Study Procedures

| Phase | Screening | Т | reatment Phas | se | Study<br>Termination |
|---|---|---|---|---|---|
| Visit Number | Visit 1[a] | Visits 2 and 3 [b] | Visit X [c] | Treatment [d] | Final Visit or<br>Early<br>Termination |
| Study Assessment | | | | | i dil |
| Obtain Informed Consent[e] | X | | | | 131 |
| Contact IRT System | X | X | X | | o X |
| Confirm Inclusion/Exclusion<br>Criteria | X | | | Š | 103 |
| Caregiver training[f] | X | X | X | Kell | |
| Medical / Surgical / Medication<br>History[g] | X | | | Mer | |
| Concomitant therapy review[g] | X | X | X | 90 | X |
| ER and EMS Visit Review [h] | | X | X | | X |
| Update PMP[i] | X | | ,iOl | | |
| Physical Examination | X[j] | X | · X | | X |
| Neurological Examination | X[j,k] | X[l] | 00, X[1] | | X[k] |
| Nasal Examination | X[j] | CAD' | X | | X |
| B-SIT | | Xaill | X | | X |
| Pregnancy Test – Urine[m] | X | XV | X | | X |
| Clinical Laboratory Testing[n] | X | X | X | | X |
| Height | X | | | | X |
| Body weight | X | X | X | | X |
| Vital Sign measurements[o] | X | X | X | | X |
| Study drug administration | 1100 | | | X | |
| Caregiver call to study center | () | | | X | |
| Record seizure activity for 24 hours after study drug administration in the subject workbook | | | | X[p] | |
| Evaluate subject's return to baseline functionality[q] | | | | X | |
| Caregiver-recorded respiration rate[r] | | | | X | |
| C-SSRS[s] | X | X | X | | X |
| Outcome questionnaires[t] | X | X | X | | X |
| Dispense Study Materials<br>Kit[u] | X[v] | | | | |
| Study Drug Kit [v] | | X | X | | |
| Drug Accountability | | X | X | | X |
| Collect and review Subject<br>Workbook | | X | X | | X |
| AE Assessment | X | X | X | X | X |

| Telephone Follow-Up [w] | Approximately every 30 days (between visits that are at least 30 days apart) |
|---|---|
|---|---|

- [a] Procedures at Visit 1 may occur at the same time as Visit 4 of the preceding double-blind study (P261-401) or up to 28 days after Visit 4 of study P261-401. If Visit 1 of this study (P261-402) is on the same day as Visit 4 of study P261-401, the procedures performed at Visit 4 of study P261-401 that are common to Visit 1 will be used for both studies. If Visit 1 for this study (P261-402) is not on the same day as Visit 4 of P261-401, all necessary procedures will be repeated, except for physical exam, neurological exam, nasal exam, and clinical laboratory testing (hematology, serum chemistry and urinalysis).
- [b] Visits 2 and 3 will take place within 120 hours (5 days) following each of the first 2 USL261-treated seizure episodes.
- [c] After Visit 3, each subject will return to the study center for a visit after every second USL261-treated episode. There is no limit on the number of seizure cluster episodes treated.
- [d] These assessments are to be completed by the caregiver(s) outside of the study center.
- [e] Informed consent provided by the subject (or subject's LAR) and caregiver before any other study specific procedures; assent may also be required for some subjects and subjects with LARs (see protocol Section 5.4 informed consent).
- [f] Caregiver training for P261-402 is required before study drug is dispensed at Visit 1. Review and re-instruct subjects and caregivers on the information provided in the training at all subsequent visits, except Final Visit or Early Termination Visit. Caregivers are also required to have a current CPR training certificate throughout the entire study.
- [g] Update from Study P261-401.
- [h] Collect number of calls to EMS and ER visits for a seizure cluster or other seizure emergency since last visit or follow-up phone call
- [i] PMP from P261-401 will be updated for this study (see protocol Section 9.3.1). PMP updates should be completed before a subject receives the study materials kit at Visit 1.
- [j] The physical, nasal, and neurological examinations performed at Visit 4 of Study P261-401 will be used for Visit 1 of this study.
- [k] Complete neurological examination.
- [1] Brief neurological examination.
- [m] Pregnancy tests required only for females of childbeating potential as described in protocol Section 6.2.2.4.
- [n]Hematology, serum chemistry, and urinalysis for all subjects; phenobarbital screen/levels for subjects taking phenobarbital and in subjects for which the investigator deems it necessary.
- [o] Blood pressure (BP), heart rate (HR), respiration rate, and body temperature.
- [p] For the first 2 years of participation in the study the date, start, and stop time of each seizure within 24 hours after any study drug administration will be recorded. After the first 2 years participation in the study, the date and start time of next seizure within 10 minutes to 24 hours after administration of the first and second dose of study drug will be recorded.
- [q] Caregiver will evaluate the subject's return to baseline functionality after each treated seizure cluster episode and record the time when the subject was able to return to what he/she was doing.
- [r]Caregiver counts the number of breaths taken by the subject during a 30-second interval. Caregivers will measure respiration rate at approximately 10, 15 and 30 minutes and 1, 2, and 4 hours after USL261 administration (see protocol Section 6.1.3).
- [s] The Since Last Visit version is administered at all visits.
- [t] The outcome questionnaires SF-12v2, TSQM, ITIQ and Caregiver Questionnaire are optional (see protocol Section 6.2.3)
- [u] The study materials kit will include at a minimum: Individualized PMP, summary of the PMP, Subject Workbook (used for collecting and recording seizure activity information, study drug administration, respiration rate, and other observations made by the caregiver), study drug kit, and dosing instructions.
- [v] One study drug kit will be dispensed at Visit 1 and Visit 2. Two study drug kits will be dispensed at Visit 3 and each Visit X
- [w] After Visit 1, telephone follow-up calls with the caregiver(s) and subject (if subject is able to communicate adequately as determined by the investigator) are to occur at least once each month (every 30 days) between visits that are at least 1 month apart until the subject has completed or prematurely discontinued from the study.

Abbreviations: B-SIT = Brief Smell Identification Test; BP = blood pressure; C-SSRS = Columbia-Suicide Severity Rating Scale; HR = heart rate; IRT = Interactive Response Technology system; LAR = legally acceptable representative; PMP = Patient Management Plan; TSQM = Treatment Satisfaction Questionnaire for Medication; ITIQ = Intranasal Therapy Impact Questionnaire

#### 3. STUDY OBJECTIVES AND CLINICAL ENDPOINTS

The study objectives are to evaluate the long-term safety and tolerability of USL-261 in the treatment of seizure clusters using the following safety endpoints:

• Caregiver-recorded respiration rate at any hour 2.1

- hour, 2 hours and 4 hours after study drug administration
- Adverse events (AEs)
- Clinical laboratory tests
- Physical, nasal, and neurological examinations
- Vital sign measurements (systolic and diastolic blood pressure, pulse rate, respiration rate, and temperature) as recorded by the study center personnel
- Brief Smell Identification Test (B-SIT)
- Columbia-Suicide Severity Rating Scale (C-SSRS)
- Requirement for unscheduled emergency room (ER) or emergency medical service (EMS) visits within 24 hours after study drug administration

### 3.2. **Clinical Endpoints**

#### 3.2.1. **Safety Endpoints**

The safety endpoints are listed above under Section 3.1, study objectives.

#### Efficacy Endpoints 3.2.2.

- Treatment Success (defined in Section 6.7.1)
- Time to return to full baseline functionality (as determined by the caregiver)

#### **Exploratory Efficacy Endpoints** 3.2.3.

- Proportion of subjects with recurrence of seizure(s) beginning 10 minutes after study drug administration to 4 hours after study drug administration
  - Time to next seizure with a start time >10 minutes after study drug administration
- Proportion of subjects with recurrence of seizure(s) beginning 10 minutes after study drug administration to 24 hours after study drug administration
- Time from administration of the first open-label dose of study drug to the second open-label dose of study drug (for subjects receiving the second dose)

#### 3.2.4. **Outcome Endpoints**

- SF-12v2 Health Survey (SF-12v2) •
- Treatment Satisfaction Questionnaire for Medication (TSQM)
- Intranasal Therapy Impact Questionnaire (ITIQ)
- Caregiver Questionnaire

#### 4. ANALYSIS POPULATIONS

#### 4.1. **Enrolled Population**

tensions or variations thereof. The Enrolled Population includes subjects who completed study P261-401, or if Study P261-401 had been terminated, also subjects who completed the Test Dose Visit (Visit 2) of Study P261-401 will also be eligible to enter this study (P261-402). All subjects must meet all the eligibility criteria in P261-402.

#### 4.2. **Safety Population**

The Safety Population includes all subjects who are enrolled in this open-label study (P261-402) and received at least one dose of open-label study drug during this open-label study (P261-402).

#### 4.3. **Efficacy Evaluable Population**

The Efficacy Evaluable Population includes all subjects in the Safety Population who have any posttreatment efficacy assessment in Study R261-402.

### GENERAL STATISTICAL CONSIDERATIONS 5.

#### 5.1. **General Consideration**

All datasets and output will be produced using SAS® Version 9.2 or higher (SAS Institute, Inc., Cary, North Carolina, USA).

### Baseline 5.2.

This study (P261-402) serves as an open-label extension for subjects who have completed study P261-401, or at least completed the test dose, if study P261-401 is terminated. The data presentations for study P261-402 will include, but are not limited to, summary of the change from baseline for the continuous safety endpoints and the outcome questionnaires (when applicable). In order to facilitate data summarization relative to exposure to active study medication, baseline endpoints will be defined as the latest non-missing value prior to Test Dose administration of USL261 from Study P261-401. Detailed baseline definitions of each endpoint of interest are presented in Table 2.

**Table 2** Baseline Definitions

| Endpoint | Baseline defined as: |
|---|---|
| Efficacy | Data displays not dependent on defining baseline |
| Vital Signs | idio |
| Weight | The last non-missing value prior to the first dose of study drug administration at Visit 2 in study |
| Laboratory Parameters | P261-401 (note the data displays for ITIQ and Caregiver Questionnaire are not dependent on |
| B-SIT | defining baseline) |
| Outcome Questionnaires (SF12-V2, TSQM) | dand |
| Physical Exam | ionally |
| Neurological Exam | D. A. I. dicatie |
| Nasal Exam | Data displays not dependent on defining baseline |
| AEs/SAEs | Data displays not dependent on defining baseline |
| C-SSRS | |

# 5.3. Handling of Missing Data

Any specific imputation procedures for missing or incomplete data will be discussed in the section describing analytic or summary methods for the corresponding variable in question. Unless otherwise stated, observed data will be presented in tables and listings without imputation of missing values.

AEs with missing start dates will be considered treatment-emergent if the stop date has been recorded and is after the first dose date (first dose date refers to the first treatment with active study drug during study P261-402).

Missing AE relationship will be presented as 'related' in tables and as missing in listings. Missing AE intensity will be considered as 'severe' in tables but will be reported as missing in listings.

# 5.4. Interim Analysis

Although no interim analysis is planned for decision making regarding this study, a snapshot of the data contained in the clinical database will be taken at the appropriate times in order for the safety data accrued in this study to be included in any regulatory submissions for this compound.

#### 5.5. Data and Safety Monitoring Board (DSMB)

The DSMB constituted for the P261-401 study will have access to the data from this study, if requested Details of the DSMB membership, meeting schedule, and data review and analysis will be documented in the DSMB Charter for the P261-401 study.

5.6. Multiple Care

#### 5.6. **Multiple Comparisons and Multiplicity**

Since this is an open-label extension study, there is no formal hypothesis testing. Where 95% confidence intervals are presented, there is no adjustment for multiple times of testing.

#### STATISTICAL ANALYSIS 6.

All analyses will be descriptive with p-values presented for the change from baseline for selected outcome assessments.

Data will be listed and tabulated overall. Continuous variables, including the change from baseline (when appropriate), will be summarized using descriptive statistics [n, mean, standard deviation (SD), minimum, median, maximum]. Categorical variables will be summarized using counts and percentages. Time to event variables will be summarized using Kaplan-Meier estimates.

Baseline is defined in Section 5.2 above, or if not included in 5.2, as the last data point prior to the first dose of study P261-402 open-label study drug administration, unless otherwise stated.

Data listings will include all subjects with at least one applicable value. Listings will be sorted by site, subject number, and date/time (if applicable).

### **Subject Disposition** 6.1.

Individual subject disposition data will be listed by investigator site for the enrolled population.

A summary of subject disposition will display the number of subjects who completed study P261-401 and were screened for the open-label study P261-402, enrolled in the open-label study P261-402, and received open-label study drug. The number of subjects who discontinued study participation will be summarized according to the primary reason for early withdrawal.

### **Treatment Exposure and Treated Seizure Clusters** 6.2.

Treatment exposure will include exposure to USL261 in study P261-402. Exposure to active study treatment will be summarized descriptively by the total number of milligrams of USL261 received per subject. Exposure data (comparative dose assignment and open-label dose usage) from study P261-401 will only be presented in listing.

The total number of seizure cluster episodes treated with USL261 will be summarized descriptively as well as categorically (number of single 5.0 mg dose [no second 5.0 mg dose] administrations of USL261, number of repeat [5.0 mg + 5.0 mg] administrations of USL261, number of total 5.0 mg administrations of USL261). For the total number of seizure cluster episodes less than or equal to 5,

categorical variables will be summarized as 1, 2 - 3, 4 - 5. For the total number of seizure cluster episodes greater than 5, categorical variables will be summarized in groups of 5, i.e. 6 - 10, 11 - 15, 16 - 20 and so on, until the maximum number based on the data.

The time on study (number of days from informed consent to the last completion / early termination visit) in study P261-402 will be summarized descriptively as well as categorically (0 - 6 months, 6 - 12 months, 12 - 24 months).

The frequency of treated seizure clusters (average per year) will be summarized descriptively as well as categorically (<2 years, 2 - <4 years, 4 - <12 years, 12 - <26 years, 26 - <52 years, >52 years).

The time between successive treated seizure clusters will be summarized descriptively as well as categorically (<=7 days, >7 - <=14 days, >14 - <=30 days, >30 - <=90 days, >90 - <=180 days, >180 days).

### **6.3.** Protocol Deviations

All instances of protocol non-compliance in study P261-402 will be tracked during the study and CSR reportable protocol deviations will be finalized by a Sponsor review prior to database lock. Protocol deviation categories will be presented in a data listing and summarized using counts and percentages. Deviations that may materially affect the evaluation of efficacy or safety will be identified as CSR Reportable. CSR Reportable protocol deviations may include, but are not limited to:

- Failure to obtain informed consent
- Failure to report a Serious Adverse Event (SAE)
- Enrolling patients outside of inclusion/exclusion criteria
- Drug dispensing/dosing errors

# **6.4.** Demographics and Baseline Characteristics

Demographics and baseline characteristics for subjects continuing in this P261-402 open-label extension study (unless otherwise specified, based on the data as collected in the preceding P261-401 study) will be presented for the Enrolled, Safety and Efficacy Evaluable Populations. Subject demographics include age (calculated as the integer number of years between date of birth and informed consent date of P261-402), age group, gender, race, ethnicity, clinical site region, height, weight, weight category, BMI, BMI category, and inducer status (based on AED exposure in P261-402). Weight recorded in pounds will be converted to kilograms and height recorded in inches will be converted to centimeters. BMI will be calculated based on weight and height using below formula:

 $BMI (kg/cm^2) = Weight/Height^2$ 

In addition subject age (years) will be categorized as follows:

- < 18 years
- $\geq 18 < 65 \text{ years}$
- $\geq$  65 years

Subject baseline characteristics include: IQ (if available), developmentally delayed status, EEG history, CT scan and/or MRI history, previous and current seizure types, seizure etiology including primary cause of epilepsy, and seizure cluster episode history.

### 6.5. Medical and Surgical History

Updates to medical and surgical history after the end of P261-401 study will be collected. Medical and surgical history will be coded using the MedDRA coding dictionary version 16.1. SOC will be sorted alphabetically and then preferred term will be sorted in order of frequency of the total column within each SOC. At each level of summarization, a subject will be counted only once for each medical and surgical history he/she has within that level. Subject listings of coded medical history terms will be provided.

### 6.6. Prior and Concomitant Medications

Prior medications are defined as medications in study P261-401 and P261-402 which started prior to the inform consent date in study P261-402. Concomitant drug therapy will include all medications (prescription or non-prescription), nutritional supplement, herbal preparation or devices (e.g., VNS) in study P261-401 and P261-402 taken/used from the inform consent date in the P261-402 open-label study through the Final Visit or ET Visit, including any with missing stop dates (or with partial missing stop dates that allow for the possibility the medication was taken after the inform consent date in study P261-402).

The World Health Organization Drug Dictionary (WHO Drug) of version December 2011 will be used to classify prior and concomitant by therapeutic class and preferred name based on ATC code level 4.

Concomitant medications will be summarized for the Safety population. Levels of summarization will include global, WHO Anatomic Therapeutic Chemical (ATC) Classification System level 3 drug class, ATC level 4 drug class, and WHO preferred name.

At each level of summarization, a subject will be counted only once for each concurrent medication he/she has within that level. The percentage of subjects having had at least one medication at each level will be calculated.

Concomitant medications excluding AEDs, prior AEDs, concomitant AEDs used for epilepsy, and concomitant AEDs used for indications other than epilepsy will be summarized separately and similar to all concomita6nt medications.

Both Prior and Concomitant AEDs will be further broken down into enzyme-inducing and non-inducing AEDs.

Separate listings will be provided for all medications and AEDs for all subjects, with medications classified as prior flagged in the listings. AEDs collected from AED page on CRF will be presumed to have 'Epilepsy' as indication. AEDs collected from concomitant medication page will be listed by indication captured on CRF.

#### 6.7. **Analyses of Efficacy and Outcome Endpoints**

Lifticacy Endpoint
All analyses of the efficacy endpoints will be conducted for the Efficacy Evaluable Population of Success

Treatment Success is a composite measure of the following criteria. Information recorded by the caregiver in the Subject Workbook will be used for analysis of the

- Termination of seizure(s) within 10 minutes after study drug administration, and
- No recurrence of seizure(s) beginning 10 minutes after study drug administration to 6 hours after study drug administration.

### 6.7.1.1.1. Derivation of Treatment Success Endpoint

Treatment Success will be determined based on data reported in the CRFs and derived programmatically for each treated seizure cluster. There are three components to be assessed in the programmatic derivation:

- 1. Termination of seizure(s) within 10 minutes. The initial seizure stopped within (≤) 10 minutes from the time of dosing and any subsequent seizures also stopped within 10 minutes of dosing.
- 2. No recurrence of seizure(s) beginning 10 minutes after study drug administration to 6 hours after study drug administration. The times of reported seizures will be used to assess if there are any seizures with start time from > 10 minutes up to  $(\leq)$  6 hours after the first dose of study drug.
- 3. No second dose given within 6 hours of the first dose of study drug administration as receiving the second dose within  $(\leq)$  6 hours confounds the efficacy evaluation of the first dose.

For each treated seizure cluster, subjects who meet all three of these components will be defined as a "Treatment Success" for that seizure cluster. If a subject does not meet all three of these components, (which may or may not be due to missing data), they will be defined as "Not a Treatment Success" for that particular seizure cluster. As subjects may be treated for multiple seizure clusters, it is possible they could meet the criteria for "Treatment Success" for some seizure clusters, but not for all.

Possible scenarios for seizure data start and stop times within the 6 hour period following the first dose of study drug are displayed below, along with the treatment success endpoint derivation (assuming no second dose was given):



The percentage of subjects achieving Treatment Success and its components (seizure termination and recurrence) will be summarized for each USL261-treated seizure cluster (first, second, etc.). Additionally, all treated seizure clusters will be pooled (across all subjects) with the proportion of Treatment Successes (this data presentation may be broken down by the number of within-subject treated seizure clusters, based on the data observed; for example, presented by subjects treated for 1-2 seizure clusters, 2-5 clusters, 3-10 clusters, etc.). Descriptive statistics for the percentage of each subject's USL261-treated seizure clusters that met the criteria for Treatment Success will also be presented.

### 6.7.1.2. Time to Return to Full Baseline Functionality (as Determined by the Caregiver)

Time to return to full baseline functionality after study P261-402 open-label study drug administration will be summarized and plotted using Kaplan-Meier estimates for each successive seizure episode (first, second, etc.) and also pooled across all treated seizure clusters. Subjects who have no records on time of return to baseline functionality within 24 hours of study drug administration and have not been administered the 2<sup>nd</sup> dose of study drug will be censored at the end of the observation period. For each seizure cluster episode, subjects who were administered the 2<sup>nd</sup> dose of open-label study drug prior to returning to baseline functionality will be censored at the time that the 2<sup>nd</sup> open-label dose was administered.

#### **6.7.2. Exploratory Efficacy Endpoints**

All exploratory efficacy analyses will be based on the Efficacy Evaluable Population.

Subjects who have been administered the second dose of the study drug (ie, 5.0 mg dose of USL261) within 4 hours of the first dose for the episode will be assumed to have had a recurrent seizure proportion of subjects with recurrence of seizure(s) recorded in the discontinuation of each success. each successive seizure cluster (first, second, etc.) and also pooled across all treated seizure clusters. Subjects who do not have a seizure recorded, or whose next seizure occurs > 4 hours after study drug administration, will be counted as not having a seizure in this particular analysis

### Time to Next Seizure with a Start Time >10 Minutes after Open-label Study Drug 6.7.2.2. Administration

Kaplan-Meier estimates and plots will be used to summarize the time-to-next seizure after study P261-402 open-label study drug administration for each successive seizure episode (first, second, etc.) and also pooled across all treated seizure clusters. Subjects who do not have another seizure before the end of the 24-hour observation period, and have not been administered the second dose of open-label study drug will be censored at the end of the observation period. Subjects who have been administered the second dose of open-label study drug and did not have a seizure before the administration of the second dose will be censored at the time of the second dose administration. The time-to-next seizure percentiles (defined based on the data) with associated 95% confidence intervals (CIs) will be displayed. The probabilities of experiencing the next seizure after open-label study drug administration at each hour up to 24 hours with associated standard error and 95% confidence intervals will be presented.

### Proportion of Subjects with Recurrence of Seizure(s) Beginning 10 Minutes after 6.7.2.3. Study Drug Administration to 24 Hours after Study Drug Administration

The proportion of subjects with recurrence of seizure(s) with a start time >10 minutes and  $\le 24$  hours after study P261-402 open-label study drug administration will be summarized for each successive seizure episode (first, second, etc.) and also pooled across all treated seizure clusters. Subjects who have been administered the second dose of open-label study drug within 24 hours will be assumed to have had a seizure. Subjects who do not have a seizure recorded with a start time >10 minutes and ≤24 hours after the administration of open-label study drug will be counted as not having a seizure in this particular analysis.

### Data Presentations / Analyses When a Second Dose is Administered

Seizure cluster episodes where both the first and second (provided if the seizure cluster has not terminated within 10 minutes after initial study drug administration or if another seizure occurs between 10 minutes and 6 hours after administration of the study drug) administrations of USL261 are given are included in the following data presentations.

### 6.7.2.4.1. Treatment Success of the Second Dose of Study Drug (5.0 mg of USL261)

Treatment Success of the second dose for subjects receiving the second dose of USL261 will be presented for each successive seizure episode (first, second, etc.) and also pooled across all treated seizure clusters.

For this analysis, Treatment Success of the second dose is defined as achieving the following:

- Termination of seizure(s) within 10 minutes after the second dose of study drug (5.0 mg of USL261)
- No recurrence of seizure(s) beginning 10 minutes after administration of the second dose of study drug (ie, 5.0 mg of USL261) to 6 hours after the second dose of study drug (5.0 mg of USL261)

Subjects whose Subject Workbook indicates seizure termination within 10 minutes of the second dose and who have no seizures recorded with start time >10 minutes and ≤6 hours after the second dose of study drug will be considered a Treatment Success of the second dose. Subjects who do not meet either of these criteria will not be considered a Treatment Success of the second dose. Similar derivation rules as used for Section 6.7.1.1 Treatment Success endpoint will be used for defining Treatment Success of the second dose, with the exception of not including the rule pertaining to the second dose.

Number and percentage will be presented for Treatment Success of the second dose and each component (seizure termination and recurrence) for subjects who received two doses of study drug. The 95% CIs for the proportions will also be presented.

# 6.7.2.4.2. Time from Administration of the First Dose of Open-Label Study Drug to the 2<sup>nd</sup> Dose

For each successive seizure episode (first, second, etc.) and also pooled across all treated seizure clusters, time (in hours) from the administration of the first dose of study P261-402 open-label study drug to the  $2^{\rm nd}$  dose (provided if the seizure cluster has not terminated within 10 minutes after initial study drug administration or if another seizure occurs between 10 minutes and 6 hours after administration of the study drug) will be descriptively summarized. In addition to the total number of subjects receiving this second dose, counts of subjects receiving the second dose in specific time categories post first dose (0 to  $\leq$ 20 minutes, >20 minutes to  $\leq$ 1 hr, >1 hr) will also be presented. For each seizure cluster episode, only subjects who received both doses of open-label study drug will be included in this data presentation.

Kaplan-Meier estimates will be used to summarize the time-to-second dose for each successive seizure episode (first, second, etc.) and also pooled across all treated seizure clusters. Subjects who do not receive the second dose of study drug within 6 hours of the initial study drug administration will be censored at the end of this 6 hour period. The time-to-second dose percentiles (defined based on the data) with associated 95% CIs will be displayed. Kaplan-Meier curves by treatment group will also be presented.

Kaplan-Meier estimates will also be used to summarize the time-to-next seizure following the second dose for each successive seizure episode (first, second, etc.) and also pooled across all treated seizure clusters. Subjects who do not have another seizure before the end of the 24-hour observation period following the second dose of study drug will be censored at the end of this observation period. The

time-to-next seizure following the second dose percentiles (defined based on the data) with associated 95% CIs will be displayed. The probabilities of experiencing the next seizure following the second dose at each hour with associated standard error and 95% confidence intervals will be presented. Kaplan-Meier curves by treatment group will also be presented.

### 6.7.2.4.3. Treatment Success for all Doses of Study Drug

An analysis similar to that in Section 6.7.2.4.1 Treatment Success of the Second Dose of Study Drug will be performed including all study drug administrations (regardless of 1<sup>st</sup> dose or 2<sup>nd</sup> dose).

The subjects and caregiver outcome assessments will be summarized using the efficacy evaluable population.

#### 6.7.3.1. SF-12v2

The SF-12v2 is a 12-item questionnaire which will be administered to both the subject and caregiver at Visit 1 and Final/ET Visit in study P261-402. All summaries will be presented separately for the subject and caregiver. Eight domains make up the SF-12v2: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. In addition, the Physical Health Component Score (PHCS) and the Mental Health Component Score (MCS) will be calculated. The scores for each domain, the PHCS and the MCS range from 0 to 100, where zero indicates the lowest level of health by the scales and 100 indicates the highest level of health.<sup>4</sup>

Summary scores for PHCS and MCS for each subject will be computed using published algorithms. Each summary measure is scored and standardized using a t-score transformation, such that a higher score represents better health status, with a mean score of 50 and a standard deviation of 10 in the general population. Missing data on the SF-12v2 will be handled as follows: domain scores will not be calculated for domains in which data are missing. Subsequently, component scores in which domain scores are missing will not be calculated.

The domain and component scores will be summarized descriptively at Baseline (defined as the last data point prior to the first dose of study drug administration at Visit 2 in study P261-401) and for Visit 1 and Final/ET Visit for study P261-402. Change from baseline will be summarized at Visit 1 and Final/ET Visit for study P261-402. For each domain and component score a paired t-test will be used to assess the within-group mean change from baseline.

#### 6.7.3.2. **Treatment Satisfaction Questionnaire for Medication (TSQM)**

The TSQM is a 14-item questionnaire that will be administered to the subject. The four TSQM scale scores calculated from the questionnaire are: effectiveness, side-effects, convenience, and global satisfaction. The TSQM scale scores are computed by adding the items loading on each factor. The lowest possible score is subtracted from the composite score and divided by the greatest possible score minus the lowest possible score. This will provide a transformed score between 0 and 1 that is then multiplied by 100. If more than one item is missing from each scale, the scale will not be calculated. Calculation of each scale score is provided below.<sup>6</sup>

**Effectiveness** 

$$([Q1 + Q2 + Q3) - 3]/18) * 100$$

If one item is missing then, ([Qx + Qy - 2]/12) \* 100 where x and y = 1, 2, or 3, with x\neq y.

### Side-Effects

If O4 is 'No' then score = 100

Else, 
$$([Q5 + Q6 + Q7 + Q8 - 4]/16) * 100$$

If one item is missing then, ([Qx + Qy + Qz - 3]/12) \* 100 where x, y, and z = 5, 6, 7, or 8,  $\pm y \neq z$ .

Nience
Q10 + Q11) - 3]/18) \* 100 with  $x\neq y\neq z$ .

### Convenience

$$([Q9 + Q10 + Q11) - 3]/18) * 100$$

If one item is missing then, ([Qx + Qy - 2]/12) \* 100 where x and y = 9,10, or 11.

### Global Satisfaction

$$([Q12 + Q13 + Q14) - 3]/14) * 100$$

Satisfaction + Q13 + Q14) - 3]/14) \* 100 If one item is missing then, ([Qx + Qy - 2]/8) \* 100 where x and y = 12, 13, or 14.

The 4 scale scores will be summarized descriptively for all visits and change from baseline (baseline is defined as the last data point prior to the first dose of study drug administration at Visit 2 in study P261-401) will be summarized for all post baseline visits. For each domain and component score a paired t-test will be used to assess the within-group mean change from baseline to each post baseline visits.

## Intranasal Therapy Impact Questionnaire (ITIQ) 6.7.3.3.

The ITIO is a two item questionnaire that is completed by both the subject and caregiver at all Visits. The level of anxiety change since subject received intranasal therapy is a scale with a range from -7 to 7, and confidence about travelling having a spray the subject can take with them is a scale from 1 to 5. The change in level of anxiety and change since subject received intranasal therapy will be summarized descriptively. Counts and percentages will be used to summarize the confidence about travelling having a spray the subject can take with them at each visit.

### Caregiver's Questionnaire 6.7.3.4.

The Caregiver Questionnaire is self-administered by the primary caregiver and consists of caregiver demographics (completed at Visit 1 or if there is a change in primary caregiver during the study) and resource utilization (completed at all visits).

All caregiver's questionnaire resource utilization data collected during the study will be presented in the listings. In addition, utilization endpoints will be summarized, including all treated seizure clusters (that is, pooled), by the categories "treatment success" and "not a treatment success" as derived for each treated seizure cluster.

### 6.8. Safety Analyses

All safety analyses will be presented based on the Safety Population unless otherwise specified. 15May2017

#### 6.8.1. **Adverse Events (AEs)**

iationsthereof Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). The actual MedDRA version used will be noted in the footnote of each corresponding output. Coding includes system organ class (SOC) and preferred term (PT). All verbatim descriptions and coded terms will be listed for all AEs.

### Pre-treatment AEs

Pre-treatment AEs will be defined as any AE that was ongoing at the end of study P261-401, or that started after the completion of study P261-401, and either ended before or did not increase in severity following open label study drug administration in P261-402. Pre-treatment AEs will be presented in a listing separate from treatment-emergent AEs (TEAEs). All summaries of AEs will be based only on and any exte TEAEs, excluding pre-treatment AEs.

### *Treatment-emergent AEs (TEAEs)*

The following AEs will be defined as TEAEs:

- Any AE that begins after the first study P261-402 open-label study drug administration;
- Any AE that begins prior to the first study P261-402 open-label study drug administration and worsens in severity following open-label study drug administration;

All AEs will be listed by subject and by MedDRA SOC and PT.

The number of events and the frequency and percentage of subjects with TEAEs/SAEs will be summarized for the Safety Population. Summary tables of TEAEs and SAEs will be presented by SOC and PT. At each summary level, a subject will be counted only once for each AE he/she experienced within that level, regardless of how many occurrences of that AE that subject experienced. The percentage of subjects having had at least one TEAE/SAE at each level will be calculated. All the TEAE analyses will also be repeated for the subset of all TEAEs that started within two days of study drug administration.

Tabular summaries will include all TEAEs, TEAEs by age group (< 18 years,  $\geq$ 18 - <65 years,  $\geq$ 65 years), TEAEs by severity (mild, moderate, severe), TEAEs by relationship to study drug, TEAEs related to study drug by severity (mild, moderate, severe), TEAEs of special interest (AESIs), serious TEAEs (SAEs) with SAEs leading to permanent discontinuation and death, SAEs by severity, and SAEs by relationship to study drug. If there are any deaths while on the study, they will be presented in a listing that includes the AE leading to death, demographic data, details of study treatment, and relationship of the AE leading to death to the study drug. In addition, listings of all TEAEs, SAEs, TEAEs of special interest (AESIs), and AEs leading to discontinuation will be presented.

The following AEs of special interest (AESIs) are discussed in this section by AESI category.

- Taste and smell disorders
- Acute central respiratory depression
- Route of administration
- Depression and suicidality/self-injury
- Abuse-related AEs

Abuse-related TEAEs will be further broken out by the following categories:

- extensions or variations thereof Drug Abuse, Dependence, Withdrawal and Substance-Related Disorders, Including Diversion
- Euphoria-related Term
- **CNS** Depressant Effects
- Stimulation and Anxiety Symptoms
- Perceptual Disturbances/Psychotomimetic Effects
- Mood Disorders and Disturbances
- Mental and Cognitive Impairment

SMQs and/or a USL-defined algorithm will be used to search AESIs. Search strategies are described in Toble 2 in Table 3.

Table 3 **Search Strategy for AESI** 

| AESI category | Search Strategy |
|---|---|
| Taste and smell disorders | Modified Taste and Smell Disorders SMQ - broad |
| Acute central respiratory depression | Modified Acute Central Respiratory Depression SMQ - broad |
| Depression and Suicidality/Self-Injury | Modified Depression and Suicidality/Self-Injury SMQ – broad |
| Route of administration | USL-defined [Oral Soft Tissue Conditions HLT (Gastrointestinal Disorders SOC); Respiratory Disorders NEC (Respiratory, Thoracic and Mediastinal Disorders SOC); Upper Respiratory Tract Disorders (Exclude Infections) (Respiratory, Thoracic and Mediastinal Disorders SOC)] — excluding overlapping terms with Acute Central Respiratory Depression SMQ and terms unrelated to MDZ NS's nasal route of administration, e.g., terms for conditions in the respiratory tract below the larynx or terms with defined causes |
| Abuse-related AEs | USL-defined algorithm |

Abbreviations: HLT=High Level Term; SMQ=Standardized MedDRA Queries; NEC=Not Elsewhere Classified.

Standard MedDRA Queries (SMQs) defined by the CIOMS Working Group are groupings of terms from one or more MedDRA SOCs that relate to a defined medical condition or area of interest. Modifications of SMQs will be documented. For hierarchical SMQs, the portion of the hierarchy to be used will be that part or those parts determined to be most relevant. A list of AEs in each category is presented in Appendix 2. Summary tables will be presented by SOC and preferred term.

In addition, "potentially clinically important" AESI will be presented for each category of AESI. AE which meets at least one of the following criteria is defined as a potentially clinically important AE:

- AE is an SAE
- AE led to discontinuation

- AE is severe in intensity and related to study drug
- AE required intervention and is related to study drug

In instances where a subject may have multiple TEAEs with differing levels of severity or relatedness, the most severe or most related event, respectively, will be reported for the severity and relatedness tables. For the purpose of summary, TEAEs with a reported relatedness of "Related", "Possibly Related", "Unlikely Related", or missing the relationship will be classified as related to study drug. TEAEs assessed as "Not Related" will be classified as not related to study drug. TEAEs with missing severity will be presented as severe in the tables but will be listed as missing.

### 6.8.2. Requirement for Unscheduled ER or EMS Visit

The number and percent of subjects requiring an unscheduled ER or EMS visit within 24 hours after study drug administration will be presented for each successive treated seizure cluster episode (first, second, etc.). In addition, the number of subjects requiring an unscheduled ER or EMS visit for any seizure cluster episode or other seizure emergency (treated or untreated) will be summarized (separately, for ER or EMS visit at any time, or visit within 24 hours after study drug administration). The total number of unscheduled ER or EMS visits will also be presented in a data listing.

### 6.8.3. Columbia-Suicide Severity Rating Scale (G-SSRS)

The C-SSRS is collected at all visits using the 'Since Last Visit' version.

### Suicidal Ideation

The number and percent of subjects with each of the following suicidal ideation scores will be summarized for each visit. The highest score for suicide ideation will be used for each subject by visit.

### Suicidal Ideation Scores

| Suicidal ideation | Score |
|---|---|
| Wish to be dead | 1 |
| Non-specific active suicidal thoughts | 2 |
| Active suicidal ideation with any methods (not planned) without intent to act | 3 |
| Active suicidal ideation with some intent to act, without specific plan | 4 |
| Active suicidal ideation with specific plan and intent | 5 |

Any suicidal ideation regardless of type will also be presented.

Each suicidal ideation severity rating will range from 0 (no ideation present) to 5 (active ideation with plan of intent). Descriptive statistics will be presented for suicidal ideation severity rating at each visit.

Descriptive statistics will also be presented for suicidal ideation intensity at each visit. The five intensity items (frequency, duration, controllability, deterrents, and reason for ideation) will be combined to create a total, sum score ranging between 0 and 25. If the subject did not have any suicidal ideation, the total score will be 0. If the subject had suicidal ideation and if one intensity item is missing, the total score will not be calculated.

### Suicidal Behavior

The number and percent of the following suicidal behaviors will be summarized for each visit.

- Actual attempt
- Engaged in non-suicidal self-injurious behavior
- Aborted attempt
- Interrupted attempts
- Preparatory acts or behavior
- Suicidal behavior
- Any suicidal behavior regardless of type
- Completed suicide

nsions of variations thereof. Descriptive statistics will be presented for the following suicidal behaviors for each visit.

- Number of attempts
- Aborted attempts
- Interrupted attempts

The number and percent of subjects with any suicidal ideation or behavior will be presented for each visit.

#### 6.8.4. Physical, Nasal, and Neurological Examinations

The number and percent of patients having normal and abnormal findings (clinically significant vs. not clinically significant) for each body system or assessment will be presented by visit for each of these exams.

#### 6.8.5. **Olfactory testing with Brief Smell Identification Test (B-SIT)**

Descriptive statistics for the summary score and changes from baseline for olfactory testing with B-SIT over time will be presented by visit. All B-SIT data will be presented in a listing.

### **Laboratory Parameters** 6.8.6.

Clinical laboratory parameters for serum chemistry, hematology, and urinalysis will be summarized descriptively at baseline and each study P261-402 visit. Mean and mean change from baseline values will be presented at each study visit. Change from baseline will be calculated at each post baseline visit as the value at that visit minus the baseline value. If either the baseline or post baseline visit value is missing, the observation will not be included in the change from baseline summary at that visit. Baseline's defined as the latest non-missing value prior to Test Dose administration of USL261 from Study P261-401.

Each laboratory result will be classified as low (L), normal (N), and high (H) at each visit according to the laboratory-supplied normal range. The shift from baseline (as defined in Section 5.2) will be presented.

Potentially clinically significant (PCS) laboratory abnormalities will be identified using standardized criteria in Appendix 1 prior to database lock and will be presented using counts and percentages. Additional displays of PCS may be presented.

#### **6.8.7.** Vital Signs / Weight

Vital sign measurements, including body weight, performed by study site staff will be presented using descriptive statistics. Vital signs, including systolic and diastolic blood pressure (mmHg), pulse (beats/min), respiration rate (breaths/min), and temperature (degrees Celsius [° C]), along with body weight, will be summarized descriptively at baseline and each study P261-402 visit. Change from baseline will be calculated as post-baseline measurement minus baseline measurement. If either the baseline or post-baseline value is missing, the observation will not be included in the change from baseline summary at that visit. Baseline is defined as the latest non-missing value prior to Test Dose administration of USL261 from Study P261-401.

The number of subjects meeting the following criteria will be presented by visit, and by time point:

- a change from baseline in systolic pressure  $\geq 40$  mm Hg diastolic blood pressure  $\leq 50$  mm Hg a change from baseline in diast. "

  pulse  $\geq 12^{\circ}$

- pulse > 120 beats per minute

  pulse < 50 beats per minute

  a change from baseline in pulse > 40 beats per minute

#### 6.8.8. **Caregiver-Recorded Respiration Rate**

The caregiver-recorded respiration rate will be presented using descriptive statistics at the scheduled collection times of (approximately) 10 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, and 4 hours after the first dose of study P261-402 open-label study drug for each successive seizure cluster episode (first, second, etc.). The number of subjects who have <8 and >24 breaths per minute will be presented by time point, across time points for each seize cluster, and across all treated seizure clusters.

#### DEVIATIONS FROM THE PROTOCOL SPECIFIED ANALYSIS 7.

The subjects and caregiver outcome assessments (detailed in Section 6.7.3) will be summarized using the efficacy evaluable population, instead of the safety population as specified in the protocol.

# MOCK TABLES, FIGURES, AND DATA LISTINGS

The mock TLGs will be provided in a separate document.

#### 9. REFERENCES

- 1. Cereghino JJ. Identification and treatment of acute repetitive seizures in children and adults.
- Glauser TA. Designing practical evidence-based treatment plans for children with prolonged seizures and status epilepticus. *J Child Neurol*. 2007;22:38S-46S.
   Utah Department of Health. Interpreting the SF12 2007. An Status Survey, 59/>
  ... A Status Survey, 59/>
  ... A Status Survey, 59/
  ... A Status Survey

**Appendix 1** Potentially Clinically Significant Laboratory Values

| | | Values | |
|---|---|---|---|
| Variable | Units | Low | High |
| Haematology | | | |
| Haemoglobin | g/L | < 10 | Not applicable |
| | g/L | > 2 decrease from baseline | > 2 increase above UL |
| Lymphocytes (Absolute) | $10^{9}/L$ | < 0.8 | Not applicable |
| Neutrophils (Absolute) | $10^{9}/L$ | < 1.5 | Not applicable |
| Platelet count | $10^{9}/L$ | < 75 | Not applicable |
| White blood cell (WBC) count | $10^{9}/L$ | < 3 | Not applicable |
| Serum Chemistry | | | 7 3/13 |
| Albumin | g/L | < 30 | Not applicable |
| Alkaline phosphotase (AP) | U/L | Not applicable | > 2.5xULN |
| Alanine aminotransferase (ALT) Grade 1 | U/L | Not applicable | $>$ ULN & $\leq$ 3xULN |
| Alanine aminotransferase (ALT) Grade 2 | U/L | Not applicable | $> 3xULN \& \le 5xULN$ |
| Alanine aminotransferase (ALT) Grade 3 | U/L ( | Not applicable | $> 5$ xULN & $\leq 20$ xUL |
| Alanine aminotransferase (ALT) Grade 4 | U/L | Not applicable | > 20xULN |
| Aspartate aminotransferase (AST) Grade 1 | UL W | Not applicable | $>$ ULN & $\leq$ 3xULN |
| Aspartate aminotransferase (AST) Grade 2 | W/Lo | Not applicable | $> 3xULN \& \le 5xULN$ |
| Aspartate aminotransferase (AST) Grade 3 | WE | Not applicable | $> 5$ xULN & $\leq 20$ xUL |
| Aspartate aminotransferase (AST) Grade 4 | U/L | Not applicable | > 20xULN |
| Bicarbonate | mmol/L | ≤ 15.9 | Not applicable |
| Calcium | mmol/L | < 2 | > 2.9 |
| Calcium Cholesterol (Total) Creatinine | mmol/L | Not applicable | > 7.75 |
| Creatinine | umol/L | Not applicable | > 1.5xULN |
| 1403 | umol/L | Not applicable | > 2x baseline |
| Gamma glutamyl transferase (GGT) | U/L | Not applicable | > 2.5xULN |
| Glucose | mmol/L | < 3.0 | > 8.9 |
| Phosphorus | mmol/L | < 0.8 | Not applicable |
| Potassium | mmol/L | < 3.0 | > 5.5 |
| Sodium | mmol/L | < 130 | > 150 |
| Total Bilirubin | umol/L | Not applicable | > 1.5xULN |
| Triglycerides | mmol/L | Not applicable | > 3.42 |

# Appendix 2 List of AEs of special interest

# (1) Abuse-related AEs (MedDRA Preferred Term):

| Drug Abuse, Dependence, Withdrawal and Substance- | Related Disorders, Including Diversion |
|---|---|
| Accidental death | Multiple drug overdose intentional |
| Accidental overdose | Nasal necrosis |
| Accidental poisoning | Nasal septum perforation |
| Dependence | Nasal septum ulceration |
| Drug abuser | Needle track marks |
| Drug administered at inappropriate site | Neonatal complications of substance abuse |
| Drug dependence | Overdose |
| Drug detoxification | Poisoning |
| Drug diversion | Polysubstance dependence |
| Drug tolerance | Prescription form tampering |
| Drug tolerance increased | Product tampering |
| Drug toxicity | Product used for unknown indication |
| Drug Withdrawal | Rebound effect |
| Drug withdrawal convulsions | Substance abuse |
| Drug withdrawal headache | Substance abuser |
| Drug withdrawal syndrome | Substance use |
| Intentional drug misuse | Substance-induced mood disorder |
| Intentional overdose | Substance-induced psychotic disorder |
| Multiple drug overdose | Treatment noncompliance |
| Multiple drug overdose accidental | Withdrawal Syndrome |
| Euphoria-related Terms | |
| Dizziness | Feeling drunk |
| Elevated mood | Feeling of relaxation |
| Euphoric mood | Inappropriate affect |
| Feeling abnormal | |
| CNS Depressant Effects | |
| Fatigue | Sluggishness |
| Lethargy | Somnolence |
| Sedation | Stupor |
| Stimulation and Anxiety Symptoms | |
| Agitation | Hypervigilance |

| Anxiety | Nervousness |
|---|---|
| Energy increased | Psychomotor hyperactivity |
| Feeling jittery | Restlessness |
| Perceptual Disturbances/Psychotomimetic Effects | |
| Abnormal dreams | Hallucinations, mixed |
| Acute psychosis | Hostility |
| Aggression | Hypoaesthesia |
| Alice in wonderland syndrome | Ideas of reference |
| Altered state of consciousness | Illogical thinking |
| Altered visual depth perception | Illusion |
| Anger | Incoherent |
| Communication disorder | Indifference |
| Confusional state | Jamais vu |
| Consciousness fluctuating | Loose associations |
| Déjà vu | Magical thinking |
| Delirium | Muscle rigidity |
| Delusion | Nightmare |
| Depersonalisation | Paraesthesia |
| Derailment Derealisation Disinhibition | Paranoia |
| Derealisation | Paroxysmal perceptual alteration |
| Disinhibition | Psychotic disorder |
| Disorientation | Reactive psychosis |
| Dissociation | Sensory disturbance |
| Dissociative disorder | Sensory level abnormal |
| Dissociative identity disorder | Somatic delusion |
| Dysarthria | Somatic hallucination |
| Fear | Staring |
| Flashback | Suspiciousness |
| Flight of ideas | Tangentiality |
| Formication | Thinking abnormal |
| Hallucination | Thought blocking |
| Hallucination, auditory | Thought broadcasting |
| Hallucination, olfactory | Thought insertion |
| Hallucination, synaesthetic | Thought withdrawal |

\_15May2017 33

| Affective disorder Affect lability Depressed mood Depression Emotional disorder Emotional distress Impatience Mood altered Mood swings Personality change Antisocial behaviour Apathy Mental and Cognitive Impairment Amnesia Cognitive disorder Disturbance in attention Memory impairment Ret | cial behaviour ntion-seeking behaviour igerence nted affect npulsions fusional arousal urbance in social behaviour ing of despair effect ulsive behaviour ia |
|---|---|
| Abnormal behaviour Affective disorder After Affect lability Depressed mood Blux Depression Con Emotional disorder Emotional distress Impatience Mood altered Mood swings Personality change Anhedonia Antisocial behaviour Apathy Mental and Cognitive Impairment Amnesia Cognitive disorder Disturbance in attention Mental impairment Mental impairment Age Mental impairment Ret | ntion-seeking behaviour igerence nted affect npulsions fusional arousal urbance in social behaviour ing of despair effect ulsive behaviour ia |
| Affective disorder Affect lability Depressed mood Depression Emotional disorder Emotional distress Impatience Mood altered Mood swings Personality change Anhedonia Antisocial behaviour Apathy Mental and Cognitive Impairment Amnesia Cognitive disorder Disturbance in attention Mental impairment Ret | ntion-seeking behaviour igerence nted affect npulsions fusional arousal urbance in social behaviour ing of despair effect ulsive behaviour ia |
| Affect lability Depressed mood Blu Depression Con Emotional disorder Emotional distress Diss Impatience Mood altered Mood swings Imp Personality change Anhedonia Antisocial behaviour Apathy Mental and Cognitive Impairment Amnesia Cognitive disorder Disturbance in attention Memory impairment Mental impairment Ret | igerence Inted affect Inpulsions Inpulsions Interpolation |
| Depression Con Emotional disorder Con Emotional distress Dis Impatience Fee Mood altered Fla Mood swings Imp Personality change Ma Anhedonia Pan Antisocial behaviour Pan Mental and Cognitive Impairment Amnesia Me Cognitive disorder Me Disturbance in attention Par Memory impairment Ret | ated affect apulsions fusional arousal arbance in social behaviour ing of despair effect alsive behaviour ia |
| Depression Con Emotional disorder Con Emotional distress Dis Impatience Fee Mood altered Flat Mood swings Imp Personality change Ma Anhedonia Part Antisocial behaviour Part Apathy Par Mental and Cognitive Impairment Amnesia Me Cognitive disorder Me Disturbance in attention Part Memory impairment Psy Mental impairment Ret | fusional arousal urbance in social behaviour ing of despair effect ulsive behaviour ia |
| Emotional disorder Emotional distress Impatience Mood altered Mood swings Personality change Anhedonia Antisocial behaviour Apathy Mental and Cognitive Impairment Amnesia Cognitive disorder Disturbance in attention Memory impairment Metal impairment Ret | fusional arousal urbance in social behaviour ing of despair effect ulsive behaviour |
| Emotional distress Impatience Mood altered Flat Mood swings Imp Personality change Anhedonia Antisocial behaviour Apathy Par Mental and Cognitive Impairment Amnesia Cognitive disorder Disturbance in attention Memory impairment Mental impairment Ret | urbance in social behaviour ing of despair effect ulsive behaviour |
| Impatience Fee Mood altered Flat Mood swings Imp Personality change Ma Anhedonia Pan Antisocial behaviour Par Apathy Par Mental and Cognitive Impairment Amnesia Me Cognitive disorder Me Disturbance in attention Par Memory impairment Psy Mental impairment Ret | ing of despair effect ulsive behaviour |
| Mood altered Mood swings Personality change Anhedonia Antisocial behaviour Apathy Mental and Cognitive Impairment Amnesia Cognitive disorder Disturbance in attention Memory impairment Metal impairment Ret | effect ulsive behaviour |
| Mood swings Personality change Anhedonia Par Antisocial behaviour Apathy Par Mental and Cognitive Impairment Amnesia Cognitive disorder Disturbance in attention Memory impairment Personality change Ma Ma Par Mental and Cognitive Impairment Me Par | effect ulsive behaviour |
| Personality change Ma Anhedonia Par Antisocial behaviour Par Apathy Par Mental and Cognitive Impairment Amnesia Me Cognitive disorder Me Disturbance in attention Par Memory impairment Psy Mental impairment Ret | ia jican |
| Anhedonia Par Antisocial behaviour Par Apathy Par Mental and Cognitive Impairment Amnesia Me Cognitive disorder Me Disturbance in attention Par Memory impairment Psy Mental impairment Ret | 1 0" |
| Antisocial behaviour Apathy Par Mental and Cognitive Impairment Amnesia Cognitive disorder Disturbance in attention Memory impairment Mental impairment Ret | c attack |
| Apathy Mental and Cognitive Impairment Amnesia Cognitive disorder Disturbance in attention Memory impairment Mental impairment Ret | |
| Mental and Cognitive Impairment Amnesia Me Cognitive disorder Me Disturbance in attention Par Memory impairment Psy Mental impairment Ret | c reaction |
| Amnesia Me Cognitive disorder Me Disturbance in attention Par Memory impairment Psy Mental impairment Ret | somnia |
| Memory impairment Psy Mental impairment Ret | |
| Memory impairment Psy Mental impairment Ret | tal disorder |
| Memory impairment Psy Mental impairment Ret | tal status changes |
| Memory impairment Psy Mental impairment Ret | mnesia |
| -0 | homotor retardation |
| | ograde amnesia |
| Psychomotor skills impaired Tra | sient global amnesia |
| Amnestic disorder Imp | aired driving ability |
| Anterograde amnesia Imp | aired reasoning |
| Balance disorder Dys | |
| Coordination abnormal Bra | ogia |
| Executive dysfunction Con | logia<br>lyphrenia |
| Judgement impaired | |

| | Executive dysfunction | | Confabulation | |
|---|---|---|---|---|
| | Judgement impaired | | | |
| curt | | | | |
| (2) AEs related to acute central respiratory depression: | | | | |
| Mis | System Organ Class | Preferred Term | | Lowest Level Term |
| | Acute central respiratory depression (SMQ) | | | |
| | Cardiac disorders | Cyanosis | | Acrocyanosis |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Acute central respiratory depression | on (SMQ) | |
| Cardiac disorders | Cardiac arrest | Arrest cardiac |
| Cardiac disorders | Cardiac arrest | Asystole |
| Cardiac disorders | Cardiac arrest | Asystolia |
| Cardiac disorders | Cardiac arrest | Asystolic |
| Cardiac disorders | Cyanosis | Blue lips Cardiac arrest |
| Cardiac disorders | Cardiac arrest | Cardiac arrest |
| Cardiac disorders | Cardiac arrest | Cardiac arrest transient |
| Cardiac disorders | Cardio-respiratory arrest | Cardio-respiratory arrest |
| Cardiac disorders | Cardio-respiratory arrest | Cardiopulmonary arrest |
| Cardiac disorders | Cardiac arrest | Congestive cardioplegia |
| Cardiac disorders | Cyanosis | Cyanosed |
| Cardiac disorders | Cyanosis | Cyanosis |
| Cardiac disorders | Cyanosis | Cyanosis NOS |
| Cardiac disorders | Cyanosis Cyanosis Cyanosis Cyanosis Cyanosis Cardiac artest | Cyanosis of lip |
| Cardiac disorders | Cyanosis | Cyanosis peripheral |
| Cardiac disorders | Cyanosis C 110 | Cyanotic |
| Cardiac disorders | Cardiac arrest | Heart arrest |
| Cardiac disorders | Cardiac arrest | Hypoxic arrest |
| Cardiac disorders | Cyanosis | Lips cyanosed |
| Cardiac disorders | Cyanosis | Nails cyanosed |
| Cardiac disorders | Cardiac arrest | Standstill cardiac |
| Cardiac disorders | Cardiopulmonary failure | Cardio-respiratory failure |
| Cardiac disorders | Cardio-respiratory distress | Cardio-respiratory distress |
| Cardiac disorders | Cardiopulmonary failure | Cardiopulmonary insufficiency |
| Cardiac disorders | Cardiopulmonary failure | Cardiopulmonary failure |
| Cardiac disorders | Cyanosis | Circumoral cyanosis |
| Cardiac disorders | Cyanosis | Cyanosis aggravated |
| Infections and infestations | Severe acute respiratory syndrome | Severe acute respiratory syndrome |
| Infections and infestations | Severe acute respiratory syndrome | SARS |
| Injury, poisoning and procedural complications | Respiratory fume inhalation disorder | Respiratory fume inhalation disorder NOS |
| Injury, poisoning and procedural complications | Respiratory fume inhalation disorder | Upper respiratory inflammation due to fumes and vapors |
| Injury, poisoning and procedural | Respiratory fume inhalation disorder | Upper respiratory inflammation due |

\_15May2017 35

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Acute central respiratory depression (SMQ) | | |
| complications | | to fumes and vapours |
| Injury, poisoning and procedural complications | Respiratory fume inhalation disorder | Smoke inhalation |
| Injury, poisoning and procedural complications | Respiratory fume inhalation disorder | Respiratory fume inhalation disorder |
| Injury, poisoning and procedural complications | Postoperative respiratory failure | Postoperative respiratory failure |
| Investigations | Blood gases abnormal | ABGs abnormal |
| Investigations | Blood gases abnormal | Abnormal arterial blood gases |
| Investigations | Breath sounds abnormal | Abnormal chest sounds |
| Investigations | Breath sounds abnormal | Abnormal chest sounds NOS |
| Investigations | Blood gases abnormal | Blood gases abnormal |
| Investigations | Blood gases abnormal | Blood gases NOS abnormal |
| Investigations | Blood pH abnormal | Blood pH abnormal |
| Investigations | Blood pH decreased | Blood pH decreased |
| Investigations | Breath sounds abnormal | Breath sounds decreased |
| Investigations | Respiratory rate decreased | Breathing rate slowed |
| Investigations | Respiratory rate decreased | Breathing slowed |
| Investigations | Breath sounds abnormal | Diminished lung sounds |
| Investigations | Blood pH decreased | Low pH |
| Investigations | Oxygen saturation abnormal | Oxygen saturation abnormal |
| Investigations | Oxygen saturation decreased | Oxygen saturation decreased |
| Investigations | Oxygen saturation decreased | Oxygen saturation low |
| Investigations | PO2 abnormal | Oxygen tension abnormal NOS |
| Investigations | PO2 decreased | Oxygen tension decreased |
| Investigations Investigations | PCO2 decreased | Partial pressure CO2 decreased |
| Investigations V | PO2 abnormal | Partial pressure O2 abnormal NOS |
| Investigations | PO2 decreased | Partial pressure O2 decreased |
| Investigations | PCO2 decreased | PCO2 decreased |
| Investigations | Blood pH decreased | pH decreased |
| Investigations | Blood pH decreased | pH reduced |
| Investigations | Blood pH decreased | Plasma pH decreased |
| Investigations | PO2 abnormal | PO2 abnormal NOS |
| Investigations | PO2 decreased | PO2 decreased |

\_15May2017 36
| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Acute central respiratory depression | on (SMQ) | |
| Investigations | PCO2 decreased | Reduced CO2 tension |
| Investigations | Respiratory rate decreased | Respiration rate decreased |
| Investigations | Respiratory rate decreased | Respiratory rate decreased |
| Investigations | Respiratory rate decreased | Respiratory rate low |
| Investigations | Breath sounds abnormal | Respiratory sounds decreased |
| Investigations | Blood pH decreased | Serum pH decreased |
| Investigations | Oxygen saturation abnormal | Oximetry abnormal |
| Investigations | Oxygen saturation decreased | Oximetry decreased |
| Investigations | Blood pH decreased | Arterial blood pH decreased |
| Investigations | Blood pH decreased | Venous blood pH decreased |
| Investigations | PCO2 abnormal | PCO2 abnormal |
| Investigations | Breath sounds abnormal | Abnormal chest sound |
| Investigations | PO2 abnormal | PO2 abnormal |
| Investigations | Breath sounds absent | Breath sounds absent |
| Investigations | Breath sounds abnormal | Breath sounds abnormal |
| Investigations | Breath sounds abnormal | Vesicular breathing abnormal |
| Investigations | Venous oxygen saturation decreased | Mixed venous blood saturation decreased |
| Investigations | Venous oxygen saturation abnormal | Mixed venous blood saturation abnormal |
| Investigations | Venous oxygen saturation decreased | SvO2 decreased |
| Investigations | Venous oxygen saturation abnormal | SvO2 abnormal |
| Investigations | Capnogram abnormal | Capnogram abnormal |
| Investigations | End-tidal CO2 abnormal | End-tidal CO2 abnormal |
| Investigations Investigations | End-tidal CO2 decreased | End-tidal CO2 decreased |
| Investigations | Alveolar oxygen partial pressure decreased | Alveolar oxygen partial pressure decreased |
| Investigations | Alveolar oxygen partial pressure abnormal | Alveolar oxygen partial pressure abnormal |
| Investigations | Venous oxygen partial pressure decreased | Venous oxygen partial pressure decreased |
| Investigations | Venous oxygen partial pressure abnormal | Venous oxygen partial pressure abnormal |
| Investigations | Venous oxygen saturation decreased | Venous oxygen saturation decreased |
| Investigations | Venous oxygen saturation abnormal | Venous oxygen saturation abnormal |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Acute central respiratory depress | ion (SMQ) | |
| Investigations | Oxygen saturation decreased | Arterial oxygen saturation decreased |
| Investigations | Oxygen saturation abnormal | Arterial oxygen saturation abnormal |
| Investigations | PO2 decreased | Arterial oxygen partial pressure decreased |
| Investigations | PO2 abnormal | Arterial oxygen partial pressure abnormal |
| Investigations | PO2 decreased | PaO2 decreased |
| Investigations | PO2 abnormal | PaO2 abnormal |
| Investigations | Breath sounds abnormal | Coarse breath sounds |
| Nervous system disorders | Central-alveolar hypoventilation | Central-alveolar hypoventilation |
| Nervous system disorders | Hypercapnic coma | Hypercapnic coma |
| Psychiatric disorders | Breath holding | Breath holding |
| Psychiatric disorders | Breath holding | Breath holding attack |
| Psychiatric disorders | Breath holding | Breath holding spells |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory distress syndrome | A.R.D.S. |
| Respiratory, thoracic and mediastinal disorders | Respiratory acidosis | Acidosis respiratory |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory failure | Acute on chronic respiratory failure |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory distress syndrome | Acute respiratory distress syndrome |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory failure | Acute respiratory failure |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory distress syndrome | Adult RDS |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory distress syndrome | Adult respiratory distress syndrome |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory distress syndrome | Adult respiratory stress syndrome |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Air hunger |
| Respiratory, thoracic and mediastinal disorders | Anoxia | Anoxia |
| Respiratory, thoracic and mediastinal disorders | Apnoea | Apnea |
| Respiratory, thoracic and mediastinal disorders | Apnoea | Apnoea |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Acute central respiratory depression | on (SMQ) | |
| Respiratory, thoracic and mediastinal disorders | Apnoeic attack | Apnoea attack |
| Respiratory, thoracic and mediastinal disorders | Apnoeic attack | Apnoeic attack |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory distress syndrome | ARDS Vall |
| Respiratory, thoracic and mediastinal disorders | Respiratory arrest | Arrest pulmonary |
| Respiratory, thoracic and mediastinal disorders | Respiratory arrest | Arrest respiratory |
| Respiratory, thoracic and mediastinal disorders | Asphyxia | Asphyxia |
| Respiratory, thoracic and mediastinal disorders | Asphyxia | Asphyxiation |
| Respiratory, thoracic and mediastinal disorders | Bradypnoea | Bradypnea |
| Respiratory, thoracic and mediastinal disorders | Bradypnoea Dyspnoea Hypopnoea | Bradypnoea |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Breath shortness |
| Respiratory, thoracic and mediastinal disorders | Hypopnoea | Breathing abnormally shallow |
| Respiratory, thoracic and mediastinal disorders | Respiratory arrest | Breathing arrested |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Breathing difficult |
| Respiratory, thoracic and mediastinal disorders | Нурорпоеа | Breathing shallow |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Breathlessness |
| Respiratory, thoracle and mediastinal disorders | Hypercapnia | Carbon dioxide narcosis |
| Respiratory, thoracic and mediastinal disorders | Sleep apnoea syndrome | Central sleep apnoea syndrome |
| Respiratory, thoracic and mediastinal disorders | Cheyne-Stokes respiration | Cheyne-Stokes respiration |
| Respiratory, thoracic and mediastinal disorders | Cyanosis central | Cyanosis central |
| Respiratory, thoracic and mediastinal disorders | Respiratory depression | Depression respiratory |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Acute central respiratory depress | ion (SMQ) | |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Difficulty breathing |
| Respiratory, thoracic and mediastinal disorders | Respiratory distress | Distress respiratory |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Dyspnea |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Dyspnea exacerbated |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Dyspnoea |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Dyspnoea exacerbated |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Dyspnoea NOS |
| Respiratory, thoracic and mediastinal disorders | Respiratory failure | Failure respiratory |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea Dyspnoea Hypercapita | Gasping |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Hunger air |
| Respiratory, thoracic and mediastinal disorders | Hypercaphia | Hypercapnia |
| Respiratory, thoracic and mediastinal disorders | Hypercaphia | Hypercapnic |
| Respiratory, thoracic and mediastinal disorders | Hypercapnia | Hypercarbia |
| Respiratory, thoracic and mediastinal disorders | Hypopnoea | Нурорпеа |
| Respiratory, thoracic and mediastinal disorders | Hypopnoea | Нурорпоеа |
| Respiratory, thoracle and mediastinal disorders | Hypoventilation | Hypoventilation |
| Respiratory, thoracic and mediastinal disorders | Нурохіа | Hypoxaemia |
| Respiratory, thoracic and mediastinal disorders | Нурохіа | Hypoxemia |
| Respiratory, thoracic and mediastinal disorders | Нурохіа | Нурохіа |
| Respiratory, thoracic and mediastinal disorders | Нурохіа | Нурохіс |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Acute central respiratory depressi | ion (SMQ) | |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Increased shortness of breath |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Increased work of breathing |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Labored breathing |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Laboured breathing |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Laboured respiration |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Marked inactivity of chest wall on inspiratory effort |
| Respiratory, thoracic and mediastinal disorders | Hypercapnia | Narcosis carbon dioxide |
| Respiratory, thoracic and mediastinal disorders | Sleep apnoea syndrome | Obstructive sleep apnoea syndrome |
| Respiratory, thoracic and mediastinal disorders | Orthopnoea Orthopnoea Orthopnoea | Orthopnea |
| Respiratory, thoracic and mediastinal disorders | Orthopnoea Chilholl | Orthopnoea |
| Respiratory, thoracic and mediastinal disorders | Respiratory arrest | Pulmonary arrest |
| Respiratory, thoracic and mediastinal disorders | Respiratory gas exchange disorder | Resp gas exchange disorder NOS |
| Respiratory, thoracic and mediastinal disorders | Respiration abnormal | Respiration abnormal |
| Respiratory, thoracic and mediastinal disorders | Cheyne-Stokes respiration | Respiration biot-type |
| Respiratory, thoracic and mediastinal disorders | Cheyne-Stokes respiration | Respiration Cheyne-Stokes-type |
| Respiratory, thoracte and mediastinal disorders | Respiratory depression | Respiration depressed |
| Respiratory, thoracic and mediastinal disorders | Respiratory failure | Respiration failure |
| Respiratory, thoracic and mediastinal disorders | Respiratory disorder | Respiration irregularity |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Respiration labored |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Respiration labored |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Acute central respiratory depress | sion (SMQ) | |
| Respiratory, thoracic and mediastinal disorders | Нурорпоеа | Respiration spontaneous decreased |
| Respiratory, thoracic and mediastinal disorders | Respiratory disorder | Respiratory abnormality, unspecified |
| Respiratory, thoracic and mediastinal disorders | Respiratory acidosis | Respiratory acidosis |
| Respiratory, thoracic and mediastinal disorders | Respiratory arrest | Respiratory arrest |
| Respiratory, thoracic and mediastinal disorders | Respiratory depression | Respiratory depression |
| Respiratory, thoracic and mediastinal disorders | Respiratory depth decreased | Respiratory depth decreased |
| Respiratory, thoracic and mediastinal disorders | Respiratory disorder | Respiratory disorder |
| Respiratory, thoracic and mediastinal disorders | Respiratory disorder | Respiratory disorder NOS |
| Respiratory, thoracic and mediastinal disorders | Respiratory distress | Respiratory distress |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory distress syndrome | Respiratory distress syndrome adult |
| Respiratory, thoracic and mediastinal disorders | Respiratory disorder | Respiratory dysfunction NOS |
| Respiratory, thoracic and mediastinal disorders | Respiratory failure | Respiratory failure |
| Respiratory, thoracic and mediastinal disorders | Respiratory gas exchange disorder | Respiratory gas exchange disorder NOS |
| Respiratory, thoracic and mediastinal disorders | Respiratory failure | Respiratory insufficiency |
| Respiratory, thoracic and mediastinal disorders | Respiratory paralysis | Respiratory paralysis |
| Respiratory, thoracle and mediastinal disorders | Respiratory disorder | Respiratory rhythm disorder |
| Respiratory, thoracic and mediastinal disorders | Respiratory disorder | Respiratory system disorder |
| Respiratory, thoracic and mediastinal disorders | Hypercapnia | Retention carbon dioxide |
| Respiratory, thoracic and mediastinal disorders | Нурорпоеа | Shallow breathing |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory distress syndrome | Shock lung |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Acute central respiratory depression | on (SMQ) | |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Short of breath |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Shortness of breath |
| Respiratory, thoracic and mediastinal disorders | Sleep apnoea syndrome | Sleep apnea |
| Respiratory, thoracic and mediastinal disorders | Sleep apnoea syndrome | Sleep apnea syndrome |
| Respiratory, thoracic and mediastinal disorders | Sleep apnoea syndrome | Sleep apnoea |
| Respiratory, thoracic and mediastinal disorders | Sleep apnoea syndrome | Sleep apnoea syndrome |
| Respiratory, thoracic and mediastinal disorders | Sleep apnoea syndrome | Sleep apnoea syndromes |
| Respiratory, thoracic and mediastinal disorders | Asphyxia | Strangulation |
| Respiratory, thoracic and mediastinal disorders | Asphyxia | Suffocation |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory distress syndrome | Surfactant deficiency syndrome adult |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory distress syndrome | Syndrome adult respiratory distress |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory distress syndrome | Syndrome respiratory distress adult |
| Respiratory, thoracic and mediastinal disorders | Respiratory disorder | Unspecified disease of respiratory system |
| Respiratory, thoracic and mediastinal disorders | Hypoventilation | Ventilation difficult |
| Respiratory, thoracic and mediastinal disorders | Respiratory failure | Ventilatory failure |
| Respiratory, thoracle and mediastinal disorders | Respiration abnormal | Respiratory sighs |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory failure | Acute respiratory decompensation |
| Respiratory, thoracic and mediastinal disorders | Respiration abnormal | Respiration abnormal NOS |
| Respiratory, thoracic and mediastinal disorders | Respiratory failure | Pulmonary failure |
| Respiratory, thoracic and mediastinal disorders | Asphyxia | Injury asphyxiation |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Acute central respiratory depress | ion (SMQ) | |
| Respiratory, thoracic and mediastinal disorders | Sleep apnoea syndrome | Apnoea syndrome |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Labored respiration |
| Respiratory, thoracic and mediastinal disorders | Apnoeic attack | Apnea attack |
| Respiratory, thoracic and mediastinal disorders | Sleep apnoea syndrome | Apnea syndrome |
| Respiratory, thoracic and mediastinal disorders | Sleep apnoea syndrome | Central sleep apnea syndrome |
| Respiratory, thoracic and mediastinal disorders | Sleep apnoea syndrome | Obstructive sleep apnea syndrome |
| Respiratory, thoracic and mediastinal disorders | Orthopnoea | Supine dyspnea |
| Respiratory, thoracic and mediastinal disorders | Orthopnoea | Supine dyspnea |
| Respiratory, thoracic and mediastinal disorders | Respiratory failure | Hypercapnic respiratory failure |
| Respiratory, thoracic and mediastinal disorders | Respiratory gas exchange disorder | Respiratory gas exchange disorder |
| Respiratory, thoracic and mediastinal disorders | Respiratory failure | Restrictive respiratory insufficiency |
| Respiratory, thoracic and mediastinal disorders | Apnoeicattack | Apneic attack |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Acute dyspnea |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Acute dyspnea |
| Respiratory, thoracic and mediastinal disorders | Cyanosis central | Cyanosis central aggravated |
| Respiratory, thoracle and mediastinal disorders | Respiratory failure | Respiratory failure aggravated |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory failure | Acute respiratory insufficiency |
| Respiratory, thoracic and mediastinal disorders | Sleep apnoea syndrome | Hypopnea syndrome |
| Respiratory, thoracic and mediastinal disorders | Sleep apnoea syndrome | Hypopnoea syndrome |
| Respiratory, thoracic and mediastinal disorders | Hypoventilation | Alveolar hypoventilation |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Acute central respiratory depression (SMQ) | | |
| Surgical and medical procedures | Oxygen supplementation | Oxygen supplementation |

## (3) AEs related to route of administration:

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration : Oral Sof | t Tissue Conditions (HLT) | e ox |
| Gastrointestinal disorders | Angina bullosa haemorrhagica | Angina bullosa haemorrhagica |
| Gastrointestinal disorders | Angina bullosa haemorrhagica | Angina bullosa hemorrhagica |
| Gastrointestinal disorders | Aphthous stomatitis | Aphthous stoma |
| Gastrointestinal disorders | Aphthous stomatitis | Aphthous stomatitis |
| Gastrointestinal disorders | Aphthous stomatitis | Aphthous ulcer |
| Gastrointestinal disorders | Aphthous stomatitis | Buccal mucosa aphthous ulceration |
| Gastrointestinal disorders | Aphthous stomatitis | Canker sores oral |
| Gastrointestinal disorders | Aphthous stomatitis | Oral aphthae |
| Gastrointestinal disorders | Aphthous stomatitis Aphthous stomatitis Aphthous stomatitis | Stomatitis aphthous |
| Gastrointestinal disorders | Aphthous stomatitis | Stomatitis ulcerative aphthous |
| Gastrointestinal disorders | Aphthous stomatitis | Ulcer aphthous |
| Gastrointestinal disorders | Aphthous stomatitis | Ulcer aphthous oral |
| Gastrointestinal disorders | Aphthous stomatitis | Ulcers aphthous oral |
| Gastrointestinal disorders | Aphthous stomatitis | Canker sore lip |
| Gastrointestinal disorders | Aphthous stomatitis | Aphthous ulcer recurrent |
| Gastrointestinal disorders | Aphthous stomatitis | Aphtha |
| Gastrointestinal disorders | Buccal mucosal roughening | Roughness oral |
| Gastrointestinal disorders | Buccal mucosal roughening | Buccal mucosal roughening |
| Gastrointestinal disorders | Buccal mucosal roughening | Rough mouth |
| Gastrointestinal disorders | Burning mouth syndrome | Burning mouth syndrome |
| Gastrointestinal disorders | Chapped lips | Lip rough |
| Gastrointesonal disorders | Chapped lips | Chapped lips |
| Gastrointestinal disorders | Chapped lips | Cracked lips |
| Gastrointestinal disorders | Cheilitis | Angular cheilitis |
| Gastrointestinal disorders | Cheilitis | Angular stomatitis |
| Gastrointestinal disorders | Cheilitis | Cheilitis |
| Gastrointestinal disorders | Cheilitis | Lip redness |
| Gastrointestinal disorders | Cheilitis | Desquamative cheilitis |
| 15May2017 | · | 45 |

15May2017 45

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration : Oral Soft | t Tissue Conditions (HLT) | |
| Gastrointestinal disorders | Cheilitis | Rash lips |
| Gastrointestinal disorders | Cheilitis | Irritation lips |
| Gastrointestinal disorders | Cheilitis | Raw lips |
| Gastrointestinal disorders | Cheilitis | Redness corner of mouth |
| Gastrointestinal disorders | Cheilitis | Inflammation lips |
| Gastrointestinal disorders | Cheilitis | Soreness corner mouth |
| Gastrointestinal disorders | Cheilitis | Sores lip |
| Gastrointestinal disorders | Cheilitis | Perleche |
| Gastrointestinal disorders | Cheilitis | Angular cheilosis |
| Gastrointestinal disorders | Cheilitis granulomatosa | Cheilitis granulomatosa |
| Gastrointestinal disorders | Cheilosis | Cheilosis |
| Gastrointestinal disorders | Contact stomatitis | Contact stomatitis |
| Gastrointestinal disorders | Enlarged uvula | Enlarged uvula |
| Gastrointestinal disorders | Gingival blister Gingival oedema | Gingival blister |
| Gastrointestinal disorders | Gingival blister | Blisters gum |
| Gastrointestinal disorders | Gingival oedema | Gingival oedema |
| Gastrointestinal disorders | Gingival codema | Oedema gum |
| Gastrointestinal disorders | Gingival oedema | Gingival edema |
| Gastrointestinal disorders | Gingival oedema | Edema gum |
| Gastrointestinal disorders | Gingival pruritus | Gingival pruritus |
| Gastrointestinal disorders | Gingival pruritus | Itching gum |
| Gastrointestinal disorders | Gingival swelling | Gingival swelling |
| Gastrointestinal disorders | Gingival swelling | Gum swelling |
| Gastrointestinal disorders | Hypoaesthesia oral | Anaesthesia lip |
| Gastrointestinal disorders | Hypoaesthesia oral | Anaesthesia mouth |
| Gastrointestinal disorders | Hypoaesthesia oral | Anaesthesia oral mucosa |
| Gastrointestinal disorders | Hypoaesthesia oral | Anaesthesia tongue |
| Gastrointestinal disorders | Hypoaesthesia oral | Hypoaesthesia oral NOS |
| Gastrointestinal disorders | Hypoaesthesia oral | Hypoaesthesia tongue |
| Gastrointestinal disorders | Hypoaesthesia oral | Numbness circumoral |
| Gastrointestinal disorders | Hypoaesthesia oral | Numbness of mouth angular |
| Gastrointestinal disorders | Hypoaesthesia oral | Numbness of tongue |
| Gastrointestinal disorders | Hypoaesthesia oral | Numbness oral |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration : Oral S | oft Tissue Conditions (HLT) | |
| Gastrointestinal disorders | Hypoaesthesia oral | Numbness perioral |
| Gastrointestinal disorders | Hypoaesthesia oral | Oral mucosal anaesthesia |
| Gastrointestinal disorders | Hypoaesthesia oral | Perioral numbness |
| Gastrointestinal disorders | Hypoaesthesia oral | Tongue sensation loss of |
| Gastrointestinal disorders | Hypoaesthesia oral | Tongue tip numbness of |
| Gastrointestinal disorders | Hypoaesthesia oral | Hypoaesthesia lips |
| Gastrointestinal disorders | Hypoaesthesia oral | Hypoaesthesia gingivat |
| Gastrointestinal disorders | Hypoaesthesia oral | Numbness mouth |
| Gastrointestinal disorders | Hypoaesthesia oral | Numb mouth |
| Gastrointestinal disorders | Hypoaesthesia oral | Numb lips |
| Gastrointestinal disorders | Hypoaesthesia oral | Numbness lips |
| Gastrointestinal disorders | Hypoaesthesia oral | Hypoaesthesia gum |
| Gastrointestinal disorders | Hypoaesthesia oral | Numbness gum |
| Gastrointestinal disorders | Hypoaesthesia oral | Numbness gingival |
| Gastrointestinal disorders | Hypoaesthesia oral | Hypoesthesia gingival |
| Gastrointestinal disorders | Hypoaesthesia oral Hypoaesthesia oral Hypoaesthesia oral Hypoaesthesia oral | Hypoesthesia lips |
| Gastrointestinal disorders | Hypoaesthesia oral | Hypoesthesia oral |
| Gastrointestinal disorders | Hypoaesthesia oral | Hypoesthesia tongue |
| Gastrointestinal disorders | Hypoaesthesia oral | Hypoaesthesia oral |
| Gastrointestinal disorders | Hypoaesthesia oral | Hypoesthesia gum |
| Gastrointestinal disorders | Hypoaesthesia oral | Anesthesia lip |
| Gastrointestinal disorders | Hypoaesthesia oral | Anesthesia mouth |
| Gastrointestinal disorders | Hypoaesthesia oral | Anesthesia oral mucosa |
| Gastrointestinal disorders | Hypoaesthesia oral | Anesthesia tongue |
| Gastrointestinal disorders | Leukoplakia oral | Leukoplakia of mouth |
| Gastrointestinal disorders | Leukoplakia oral | Leukoplakia of oral mucosa, including tongue |
| Gastrointestinal disorders | Leukoplakia oral | Leukoplakia oral |
| Gastrointestinal disorders | Leukoplakia oral | Leukoplakia oral NOS |
| Gastrointestinal disorders | Leukoplakia oral | Oral leukoplakia NOS |
| Gastrointestinal disorders | Leukoplakia oral | Leukoplakia buccalis |
| Gastrointestinal disorders | Leukoplakia oral | Leukoplakia labialis |
| Gastrointestinal disorders | Leukoplakia oral | Leukoplakia lingualis |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration : Oral So | ft Tissue Conditions (HLT) | |
| Gastrointestinal disorders | Leukoplakia oral | Leukoplakia of oral mucosa, incl tongue |
| Gastrointestinal disorders | Leukoplakia oral | Leukoplakia tongue |
| Gastrointestinal disorders | Lip blister | Blister of lip |
| Gastrointestinal disorders | Lip blister | Lip blister |
| Gastrointestinal disorders | Lip blister | Blister lip |
| Gastrointestinal disorders | Lip discolouration | Lip colour altered |
| Gastrointestinal disorders | Lip discolouration | Lip discolouration |
| Gastrointestinal disorders | Lip discolouration | Lip color altered |
| Gastrointestinal disorders | Lip discolouration | Lip discoloration |
| Gastrointestinal disorders | Lip disorder | Lip disorder NOS |
| Gastrointestinal disorders | Lip disorder | Lip disorder |
| Gastrointestinal disorders | Lip disorder | Bumps lip |
| Gastrointestinal disorders | Lip erosion Lip exfoliation Lip exfoliation Lip exfoliation | Lip erosion |
| Gastrointestinal disorders | Lip exfoliation | Lip sloughing |
| Gastrointestinal disorders | Lip exfoliation | Peeling lips |
| Gastrointestinal disorders | Lip exfoliation | Lip exfoliation |
| Gastrointestinal disorders | Lip haematoma | Lip haematoma |
| Gastrointestinal disorders | Lip haematoma | Lip hematoma |
| Gastrointestinal disorders | Lip haemorrhage | Lip haemorrhage |
| Gastrointestinal disorders | Lip haemorrhage | Hemorrhage lips |
| Gastrointestinal disorders | Lip haemorrhage | Bleeding lips |
| Gastrointestinal disorders | Lip haemorrhage | Lip hemorrhage |
| Gastrointestinal disorders | Lip haemorrhage | Haemorrhage lips |
| Gastrointestinal disorders | Lip haemorrhage | Lip bleeding |
| Gastrointestinal disorders | Lip oedema | Edema lip |
| Gastrointestinal disorders | Lip oedema | Lip edema |
| Gastrointestinal disorders | Lip oedema | Lip oedema |
| Gastrointestinal disorders | Lip oedema | Oedema lip |
| Gastrointestinal disorders | Lip pain | Lip pain |
| Gastrointestinal disorders | Lip pain | Lip sore |
| Gastrointestinal disorders | Lip pain | Lip soreness |
| Gastrointestinal disorders | Lip pain | Tender lips |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration : Oral Soft | t Tissue Conditions (HLT) | |
| Gastrointestinal disorders | Lip pain | Stinging lips |
| Gastrointestinal disorders | Lip pain | Sensitive lips |
| Gastrointestinal disorders | Lip pruritus | Lip pruritus |
| Gastrointestinal disorders | Lip swelling | Lip swelling |
| Gastrointestinal disorders | Lip swelling | Lips swelling non-specific |
| Gastrointestinal disorders | Lip swelling | Swelling lips |
| Gastrointestinal disorders | Lip swelling | Swelling of lips |
| Gastrointestinal disorders | Lip swelling | Swollen lips |
| Gastrointestinal disorders | Lip ulceration | Lip ulcer |
| Gastrointestinal disorders | Lip ulceration | Lip ulceration |
| Gastrointestinal disorders | Lip ulceration | Ulcerlip |
| Gastrointestinal disorders | Melanoplakia oral | Melanoplakia oral |
| Gastrointestinal disorders | Mouth haemorrhage | Hemorrhage mouth |
| Gastrointestinal disorders | Mouth haemorrhage Mouth haemorrhage | Hemorrhage of mouth |
| Gastrointestinal disorders | Mouth haemorrhage | Hemorrhage oral |
| Gastrointestinal disorders | Mouth haemorrhage | Mouth haemorrhage |
| Gastrointestinal disorders | Mouth haemorrhage | Mouth hemorrhage |
| Gastrointestinal disorders | Mouth haemorrhage | Oral haemorrhage |
| Gastrointestinal disorders | Mouth haemorrhage | Oral hemorrhage |
| Gastrointestinal disorders | Mouth haemorrhage | Oral mucosa bleeding |
| Gastrointestinal disorders | Mouth haemorrhage | Oral mucosa ecchymosis |
| Gastrointestinal disorders | Mouth haemorrhage | Oral mucosal petechiae |
| Gastrointestinal disorders | Mouth haemorrhage | Petechiae oral mucosa |
| Gastrointestinal disorders | Mouth haemorrhage | Bleeding mouth |
| Gastrointestinal disorders | Mouth haemorrhage | Haemorrhage mouth |
| Gastrointestinal disorders | Mouth haemorrhage | Haemorrhage of mouth |
| Gastrointestinal disorders | Mouth haemorrhage | Haemorrhage oral |
| Gastrointestinal disorders | Mouth haemorrhage | Mouth bleeding |
| Gastrointestinal disorders | Mouth ulceration | Buccal mucosa ulceration |
| Gastrointestinal disorders | Mouth ulceration | Buccal ulceration |
| Gastrointestinal disorders | Mouth ulceration | Mouth ulcer |
| Gastrointestinal disorders | Mouth ulceration | Mouth ulceration |
| Gastrointestinal disorders | Mouth ulceration | Oral ulceration |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration : Oral Soft | t Tissue Conditions (HLT) | |
| Gastrointestinal disorders | Mouth ulceration | Stomatitis ulcerative |
| Gastrointestinal disorders | Mouth ulceration | Ulcer buccal |
| Gastrointestinal disorders | Mouth ulceration | Ulcer mouth |
| Gastrointestinal disorders | Mouth ulceration | Ulceration mouth |
| Gastrointestinal disorders | Mouth ulceration | Ulceration of mouth |
| Gastrointestinal disorders | Mouth ulceration | Ulcerative stomatitis |
| Gastrointestinal disorders | Mouth ulceration | Ulcerative stomatitis, acute |
| Gastrointestinal disorders | Mouth ulceration | Mouth ulceration aggravated |
| Gastrointestinal disorders | Odynophagia | Odynophagia |
| Gastrointestinal disorders | Odynophagia | Swallowing painful |
| Gastrointestinal disorders | Oedema mouth | Edema of mouth |
| Gastrointestinal disorders | Oedema mouth | Oedema mouth |
| Gastrointestinal disorders | Oedema mouth | Oral mucosa swollen |
| Gastrointestinal disorders | Oedema mouth Oedema mouth Oedema mouth Oedema mouth Oral discharge | Swollen mouth |
| Gastrointestinal disorders | Oedema mouth | Edema mouth |
| Gastrointestinal disorders | Oedema mouth | Oedema of mouth |
| Gastrointestinal disorders | Oral discharge | Oral discharge |
| Gastrointestinal disorders | Oral discomfort | Burning oral sensation |
| Gastrointestinal disorders | Oral discomfort | Discomfort in mouth |
| Gastrointestinal disorders | Oral discomfort | Lip burning sensation of |
| Gastrointestinal disorders | Oral discomfort | Oral cavity discomfort |
| Gastrointestinal disorders | Oral discomfort | Oral discomfort |
| Gastrointestinal disorders | Oral discomfort | Oral hot feeling |
| Gastrointestinal disorders | Oral discomfort | Burning corner of mouth |
| Gastrointestinal disorders | Oral discomfort | Burning lips |
| Gastrointestinal disorders | Oral discomfort | Burning mouth |
| Gastrointestinal disorders | Oral disorder | Oral soft tissue disorder NOS |
| Gastrointestinal disorders | Oral disorder | Oral mucosal disorder |
| Gastrointestinal disorders | Oral disorder | Oral lesion |
| Gastrointestinal disorders | Oral disorder | Oral soft tissue disorder |
| Gastrointestinal disorders | Oral disorder | Oral disorder |
| Gastrointestinal disorders | Oral disorder | Mouth bump |
| Gastrointestinal disorders | Oral dysaesthesia | Dysesthesia of lips |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration : Oral Soft | t Tissue Conditions (HLT) | |
| Gastrointestinal disorders | Oral dysaesthesia | Dysesthesia of tongue |
| Gastrointestinal disorders | Oral dysaesthesia | Oral dysaesthesia |
| Gastrointestinal disorders | Oral dysaesthesia | Oral dysesthesia |
| Gastrointestinal disorders | Oral dysaesthesia | Dysaesthesia of lips |
| Gastrointestinal disorders | Oral dysaesthesia | Dysaesthesia of tongue |
| Gastrointestinal disorders | Oral dysaesthesia | Dysaesthesia of tongue Vincent's symptom |
| Gastrointestinal disorders | Oral leukoedema | Oral leukoedema |
| Gastrointestinal disorders | Oral lichen planus | Oral lichen planus |
| Gastrointestinal disorders | Oral mucosa atrophy | Oral mucosa atrophy |
| Gastrointestinal disorders | Oral mucosa erosion | Oral mucosa erosion |
| Gastrointestinal disorders | Oral mucosal blistering | Blistering of mouth |
| Gastrointestinal disorders | Oral mucosal blistering | Oral mucosa blister |
| Gastrointestinal disorders | Oral mucosal blistering | Oral mucosa blistering |
| Gastrointestinal disorders | Oral mucosal blistering | Oral mucosal blistering |
| Gastrointestinal disorders | Oral mucosal discolouration | Oral mucosa discolouration |
| Gastrointestinal disorders | Oral mucosal discolouration | Oral mucosal discolouration |
| Gastrointestinal disorders | Oral mucosal discolouration | Oral mucosal discoloration |
| Gastrointestinal disorders | Oral mucosal cruption | Oral mucosal eruption |
| Gastrointestinal disorders | Oral mucosal erythema | Oral mucosa redness |
| Gastrointestinal disorders | Oral mucosal erythema | Oral redness |
| Gastrointestinal disorders | Oral mucosal erythema | Redness mouth |
| Gastrointestinal disorders | Oral mucosal erythema | Oral mucosal erythema |
| Gastrointestinal disorders | Oral mucosal erythema | Palatal erythema |
| Gastrointestinal disorders | Oral mucosal exfoliation | Oral mucosal sloughing |
| Gastrointestinal disorders | Oral mucosal exfoliation | Sloughing of buccal mucosa |
| Gastrointestinal disorders | Oral mucosal exfoliation | Sloughing of mouth |
| Gastrointestinal disorders | Oral mucosal exfoliation | Gingival sloughing |
| Gastrointestinal disorders | Oral mucosal exfoliation | Peeling mouth |
| Gastrointestinal disorders | Oral mucosal exfoliation | Desquamation mouth |
| Gastrointestinal disorders | Oral mucosal exfoliation | Sloughing gums |
| Gastrointestinal disorders | Oral mucosal exfoliation | Sloughing gingival |
| Gastrointestinal disorders | Oral mucosal exfoliation | Peeling gingival |
| Gastrointestinal disorders | Oral mucosal exfoliation | Peeling gum |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration : Oral S | oft Tissue Conditions (HLT) | |
| Gastrointestinal disorders | Oral mucosal exfoliation | Desquamation gum |
| Gastrointestinal disorders | Oral mucosal exfoliation | Desquamation gingival |
| Gastrointestinal disorders | Oral mucosal exfoliation | Oral mucosal exfoliation |
| Gastrointestinal disorders | Oral mucosal hypertrophy | Oral mucosal hypertrophy |
| Gastrointestinal disorders | Oral pain | Mouth pain |
| Gastrointestinal disorders | Oral pain | Oral angular pain |
| Gastrointestinal disorders | Oral pain | Oral mucosa pain |
| Gastrointestinal disorders | Oral pain | Oral pain |
| Gastrointestinal disorders | Oral pain | Pain mouth |
| Gastrointestinal disorders | Oral pain | Pain oral |
| Gastrointestinal disorders | Oral pain | Sore mouth |
| Gastrointestinal disorders | Oral pain | Sensitive mouth |
| Gastrointestinal disorders | Oral pain | Tender mouth |
| Gastrointestinal disorders | Oral pain Oral pain Oral pain Oral papule Oral pruritus | Stinging mouth |
| Gastrointestinal disorders | Oral pain | Soreness roof of mouth |
| Gastrointestinal disorders | Oral papule | Oral papule |
| Gastrointestinal disorders | Oral pruritus | Intraoral pruritus |
| Gastrointestinal disorders | Oral pruritus | Itching mouth |
| Gastrointestinal disorders | Oral pruntus | Oral pruritus |
| Gastrointestinal disorders | Oral submucosal fibrosis | Oral submucosal fibrosis |
| Gastrointestinal disorders | Oral submucosal fibrosis | Oral submucous fibrosis, including of tongue |
| Gastrointestinal disorders | Oral submucosal fibrosis | Oral submucous fibrosis, incl of tongue |
| Gastrointestinal disorders | Oral toxicity | Oral toxicity |
| Gastrointestinal disorders | Palatal disorder | Palatal disorder |
| Gastrointestinal disorders | Palatal disorder | Palatal lesion |
| Gastrointestinal disorders | Palatal disorder | Palatal nodule |
| Gastrointestinal disorders | Palatal disorder | Soft palate disorder |
| Gastrointestinal disorders | Palatal dysplasia | Palatal dysplasia |
| Gastrointestinal disorders | Palatal oedema | Palatine arch swollen |
| Gastrointestinal disorders | Palatal oedema | Oedema uvula |
| Gastrointestinal disorders | Palatal oedema | Edema uvula |
| Gastrointestinal disorders | Palatal oedema | Palatal oedema |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration : Oral Soft | t Tissue Conditions (HLT) | |
| Gastrointestinal disorders | Palatal oedema | Palatal edema |
| Gastrointestinal disorders | Palatitis | Palatitis |
| Gastrointestinal disorders | Paraesthesia oral | Circumoral paresthesia |
| Gastrointestinal disorders | Paraesthesia oral | Mouth paresthesia |
| Gastrointestinal disorders | Paraesthesia oral | Paraesthesia circumoral |
| Gastrointestinal disorders | Paraesthesia oral | Paraesthesia mouth |
| Gastrointestinal disorders | Paraesthesia oral | Paraesthesia oral NOS |
| Gastrointestinal disorders | Paraesthesia oral | Paraesthesia tongue |
| Gastrointestinal disorders | Paraesthesia oral | Paresthesia circumoral |
| Gastrointestinal disorders | Paraesthesia oral | Paresthesia mouth |
| Gastrointestinal disorders | Paraesthesia oral | Tongue abnormal feeling of |
| Gastrointestinal disorders | Paraesthesia oral | Paraesthesia lips |
| Gastrointestinal disorders | Paraesthesia oral | Paraesthesia gingival |
| Gastrointestinal disorders | Paraesthesia oral | Tingling mouth |
| Gastrointestinal disorders | Paraesthesia oral | Tingling lips |
| Gastrointestinal disorders | Paraesthesia oral Paraesthesia oral Paraesthesia oral Paraesthesia oral | Paresthesia lips |
| Gastrointestinal disorders | Paraesthesia oral | Tingling tongue |
| Gastrointestinal disorders | Paraesthesia oral | Tingling gum |
| Gastrointestinal disorders | Paraesthesia oral | Tingling gingival |
| Gastrointestinal disorders | Paraesthesia oral | Paraesthesia gum |
| Gastrointestinal disorders | Paraesthesia oral | Paresthesia gingival |
| Gastrointestinal disorders | Paraesthesia oral | Paresthesia gum |
| Gastrointestinal disorders | Paraesthesia oral | Paresthesia oral |
| Gastrointestinal disorders | Paraesthesia oral | Paresthesia tongue |
| Gastrointestinal disorders | Paraesthesia oral | Paraesthesia oral |
| Gastrointestinal disorders | Paraesthesia oral | Perioral tingling |
| Gastrointestinal disorders | Paraesthesia oral | Perioral paraesthesia |
| Gastrointestinal disorders | Paraesthesia oral | Perioral paresthesia |
| Gastrointestinal disorders | Pigmentation buccal | Pigmentation buccal |
| Gastrointestinal disorders | Pigmentation lip | Lip pigmental spot |
| Gastrointestinal disorders | Pigmentation lip | Lip pigmentation |
| Gastrointestinal disorders | Pigmentation lip | Pigmentation lip |
| Gastrointestinal disorders | Pyostomatitis vegetans | Pyostomatitis vegetans |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration : Oral Sof | t Tissue Conditions (HLT) | |
| Gastrointestinal disorders | Stomatitis | Buccal inflammation |
| Gastrointestinal disorders | Stomatitis | Mouth irritation |
| Gastrointestinal disorders | Stomatitis | Mucositis oral |
| Gastrointestinal disorders | Stomatitis | Stomatitis |
| Gastrointestinal disorders | Stomatitis | Sores mouth |
| Gastrointestinal disorders | Stomatitis | Sores roof of mouth |
| Gastrointestinal disorders | Stomatitis | Raw mouth |
| Gastrointestinal disorders | Stomatitis | Irritation roof of mouth |
| Gastrointestinal disorders | Stomatitis | Chapped mouth |
| Gastrointestinal disorders | Stomatitis | Inflammation of mouth |
| Gastrointestinal disorders | Stomatitis | Mouth broke out |
| Gastrointestinal disorders | Stomatitis | daflammation under tongue |
| Gastrointestinal disorders | Stomatitis | Oral mucosal irritation |
| Gastrointestinal disorders | Stomatitis | Vesicular stomatitis |
| Gastrointestinal disorders | Stomatitis | Gingivostomatitis |
| Gastrointestinal disorders | Stomatitis C 1800 | Pseudomembranous stomatitis |
| Gastrointestinal disorders | Stomatitis haemorrhagic | Stomatitis haemorrhagic |
| Gastrointestinal disorders | Stomatitis haemorrhagic | Stomatitis hemorrhagic |
| Gastrointestinal disorders | Stomatitis necrotising | Cancrum oris |
| Gastrointestinal disorders | Stomatitis necrotising | Mouth necrosis |
| Gastrointestinal disorders | Stomatitis necrotising | Necrosis mouth |
| Gastrointestinal disorders | Stomatitis necrotising | Noma |
| Gastrointestinal disorders | Stomatitis necrotising | Stomatitis necrotising |
| Gastrointestinal disorders | Stomatitis necrotising | Stomatitis necrotizing |
| Gastrointestinal disorders | Uvulitis | Uvulitis |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Respirato | ory Disorders NEC (HLT) | |
| Respiratory, thoracic and mediastinal disorders | Allergic cough | Allergic cough |
| Respiratory, thoracic and mediastinal disorders | Choking | Choked on food |
| Respiratory, thoracic and mediastinal disorders | Choking | Choking |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Respiratory Disorders NEC (HLT) | | |
| Respiratory, thoracic and mediastinal disorders | Choking | Choke on medication |
| Respiratory, thoracic and mediastinal disorders | Choking sensation | Choking sensation |
| Respiratory, thoracic and mediastinal disorders | Choking sensation | Choking sensation (excl psychogenic and dysphagia) |
| Respiratory, thoracic and mediastinal disorders | Choking sensation | Pharynx closed sensation of |
| Respiratory, thoracic and mediastinal disorders | Choking sensation | Pharynx strangled sensation of |
| Respiratory, thoracic and mediastinal disorders | Cough | Cough |
| Respiratory, thoracic and mediastinal disorders | Cough | Cough increased |
| Respiratory, thoracic and mediastinal disorders | Cough | Cough nonproductive |
| Respiratory, thoracic and mediastinal disorders | Cough Cough Cough Cough Cough Cough | Cough resembling asthma |
| Respiratory, thoracic and mediastinal disorders | Cough | Coughing |
| Respiratory, thoracic and mediastinal disorders | Cough Clind | Dry cough |
| Respiratory, thoracic and mediastinal disorders | Cough | Irritant cough |
| Respiratory, thoracic and mediastinal disorders | Cough | Irritative cough |
| Respiratory, thoracic and mediastinal disorders | Cough | Nocturnal cough |
| Respiratory, thoracic and mediastinal disorders | Cough | Persistent dry cough |
| Respiratory, thoracle and mediastinal disorders | Cough | Persistent non-productive cough |
| Respiratory, thoracic and mediastinal disorders | Cough | Cough aggravated |
| Respiratory, thoracic and mediastinal disorders | Cough | Coughing after drug inhalation |
| Respiratory, thoracic and mediastinal disorders | Cough | Drug-induced cough |
| Respiratory, thoracic and mediastinal disorders | Cough | Smoker's cough |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Respira | tory Disorders NEC (HLT) | |
| Respiratory, thoracic and mediastinal disorders | Cough | Paroxysmal cough |
| Respiratory, thoracic and mediastinal disorders | Cough | Acute cough |
| Respiratory, thoracic and mediastinal disorders | Cough | Chronic cough |
| Respiratory, thoracic and mediastinal disorders | Cough | Persistent cough |
| Respiratory, thoracic and mediastinal disorders | Cough | Painful cough |
| Respiratory, thoracic and mediastinal disorders | Cough | Cough ineffective |
| Respiratory, thoracic and mediastinal disorders | Cough | Cough weak |
| Respiratory, thoracic and mediastinal disorders | Cough decreased | Cough decreased |
| Respiratory, thoracic and mediastinal disorders | Dry throat Dry throat Dry throat | Dry throat |
| Respiratory, thoracic and mediastinal disorders | Dry throat | Pharynx dry |
| Respiratory, thoracic and mediastinal disorders | Dry throat | Throat dry |
| Respiratory, thoracic and mediastinal disorders | Dysphoma | Distorted voice |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Disturbance in loudness |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Dysphonia |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Hoarse voice |
| Respiratory, thoracie and mediastinal disorders | Dysphonia | Hoarseness |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Hoarseness of voice |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Phonation difficulty |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Resonance disorder |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Vocal tone disorder |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Respirat | tory Disorders NEC (HLT) | |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Vocal volume disorder |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Voice alteration |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Voice disturbance |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Voice disturbance, unspecified |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Voice lowered |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Hypophonia |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Rhinolalia |
| Respiratory, thoracic and mediastinal disorders | Haemoptysis | Blood streaked sputum |
| Respiratory, thoracic and mediastinal disorders | Haemoptysis Haemoptysis Haemoptysis | Coughing blood |
| Respiratory, thoracic and mediastinal disorders | Haemoptysis Chillion | Haemoptysis |
| Respiratory, thoracic and mediastinal disorders | Haemoptosis | Hemoptysis |
| Respiratory, thoracic and mediastinal disorders | Haemoptysis | Sputum bloody |
| Respiratory, thoracic and mediastinal disorders | Hiccups | Hiccough |
| Respiratory, thoracic and mediastinal disorders | Hiccups | Hiccup |
| Respiratory, thoracic and mediastinal disorders | Hiccups | Hiccups |
| Respiratory, thoracle and mediastinal disorders | Hiccups | Singultation |
| Respiratory, thoracic and mediastinal disorders | Hiccups | Singultous |
| Respiratory, thoracic and mediastinal disorders | Hiccups | Singultus |
| Respiratory, thoracic and mediastinal disorders | Hiccups | Intractable hiccups |
| Respiratory, thoracic and mediastinal disorders | Increased bronchial secretion | Airway secretion excessive |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Respiratory Disorders NEC (HLT) | | |
| Respiratory, thoracic and mediastinal disorders | Increased bronchial secretion | Bronchial secretion excessive |
| Respiratory, thoracic and mediastinal disorders | Increased bronchial secretion | Bronchorrhea |
| Respiratory, thoracic and mediastinal disorders | Increased bronchial secretion | Bronchorrhoea |
| Respiratory, thoracic and mediastinal disorders | Increased bronchial secretion | Excessive bronchial secretion |
| Respiratory, thoracic and mediastinal disorders | Increased bronchial secretion | Tracheo-bronchial secretion excess |
| Respiratory, thoracic and mediastinal disorders | Increased bronchial secretion | Increased bronchial secretion |
| Respiratory, thoracic and mediastinal disorders | Increased upper airway secretion | Throat secretion increased |
| Respiratory, thoracic and mediastinal disorders | Increased upper airway secretion | Phlegm |
| Respiratory, thoracic and mediastinal disorders | Increased upper airway secretion | Increased upper airway secretion |
| Respiratory, thoracic and mediastinal disorders | Increased viscosity of bronchial secretion | Sputum viscosity increased |
| Respiratory, thoracic and mediastinal disorders | Increased viscosity of bronchial secretion | Increased viscosity of bronchial secretion |
| Respiratory, thoracic and mediastinal disorders | Increased viscosity of nasal secretion | Increased viscosity of nasal secretion |
| Respiratory, thoracic and mediastinal disorders | Increased viscosity of nasal secretion | Thick nasal mucus |
| Respiratory, thoracic and mediastinal disorders | Laryngeal discomfort | Laryngeal discomfort |
| Respiratory, thoracic and mediastinal disorders | Laryngeal discomfort | Pharyngolaryngeal discomfort |
| Respiratory, thoracie and mediastinal disorders | Laryngeal pain | Laryngeal pain |
| Respiratory, thoracic and mediastinal disorders | Laryngeal pain | Larynx burning pain of |
| Respiratory, thoracic and mediastinal disorders | Laryngeal pain | Larynx pain |
| Respiratory, thoracic and mediastinal disorders | Laryngeal pain | Pharyngolaryngeal pain |
| Respiratory, thoracic and mediastinal disorders | Mouth breathing | Jaw breathing |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Respirat | tory Disorders NEC (HLT) | |
| Respiratory, thoracic and mediastinal disorders | Mouth breathing | Mouth breathing |
| Respiratory, thoracic and mediastinal disorders | Nasal discharge discolouration | Nasal discharge discolouration |
| Respiratory, thoracic and mediastinal disorders | Nasal discharge discolouration | Nasal discharge discoloration |
| Respiratory, thoracic and mediastinal disorders | Nasal discomfort | Discomfort in nose |
| Respiratory, thoracic and mediastinal disorders | Nasal discomfort | Nasal burning |
| Respiratory, thoracic and mediastinal disorders | Nasal discomfort | Nasal cavity strange sensation of |
| Respiratory, thoracic and mediastinal disorders | Nasal discomfort | Nasaturitation |
| Respiratory, thoracic and mediastinal disorders | Nasal discomfort | Nasal itching |
| Respiratory, thoracic and mediastinal disorders | Nasal discomfort | Nasal passage irritation |
| Respiratory, thoracic and mediastinal disorders | Nasal discomfort | Nasal soreness |
| Respiratory, thoracic and mediastinal disorders | Nasal discomfort | Sore nose |
| Respiratory, thoracic and mediastinal disorders | Nasal discomfort | Nasal discomfort |
| Respiratory, thoracic and mediastinal disorders | Nasal flaring | Nasal flaring |
| Respiratory, thoracic and mediastinal disorders | Nasal obstruction | Nasal obstruction |
| Respiratory, thoracic and mediastinal disorders | Nasal obstruction | Nasal obstruction increased |
| Respiratory, thoracte and mediastinal disorders | Nasopharyngeal reflux | Nasopharyngeal reflux |
| Respiratory, thoracic and mediastinal disorders | Nocturnal dyspnoea | Nocturnal dyspnoea |
| Respiratory, thoracic and mediastinal disorders | Nocturnal dyspnoea | Nocturnal dyspnea |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal blistering | Oropharyngeal blistering |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal discomfort | Pharynx discomfort |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Respira | atory Disorders NEC (HLT) | |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal discomfort | Pharynx ill sensation of |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal discomfort | Pharynx strange sensation of |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal discomfort | Oropharyngeal discomfort |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal pain | Pain pharynx |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal pain | Pain throat |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal pain | Sore throat |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal pain | Sore throat NOS |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal pain | Throat pain |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal pain | Throat sore |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal pain | Chronic sore throat |
| Respiratory, thoracic and mediastinal disorders | Oropharyageal pain | Oropharyngeal pain |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal plaque | Mouth plaque |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal plaque | Plaque mouth |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal plaque | Oropharyngeal plaque |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal scar | Oropharyngeal scar |
| Respiratory, thoracle and mediastinal disorders | Paranasal sinus discomfort | Paranasal sinus discomfort |
| Respiratory thoracic and mediastinal disorders | Productive cough | Productive cough |
| Respiratory, thoracic and mediastinal disorders | Productive cough | Sputum |
| Respiratory, thoracic and mediastinal disorders | Productive cough | Expectoration |
| Respiratory, thoracic and mediastinal disorders | Respiratory tract oedema | Respiratory tract oedema |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Respirat | tory Disorders NEC (HLT) | |
| Respiratory, thoracic and mediastinal disorders | Respiratory tract oedema | Airway oedema |
| Respiratory, thoracic and mediastinal disorders | Respiratory tract oedema | Airway edema |
| Respiratory, thoracic and mediastinal disorders | Respiratory tract oedema | Respiratory tract edema |
| Respiratory, thoracic and mediastinal disorders | Rhinalgia | Nasal stinging |
| Respiratory, thoracic and mediastinal disorders | Rhinalgia | Stinging of nose |
| Respiratory, thoracic and mediastinal disorders | Rhinalgia | Rhinalgia |
| Respiratory, thoracic and mediastinal disorders | Rhinalgia | Nasat pain |
| Respiratory, thoracic and mediastinal disorders | Rhinorrhoea | Nasal discharge |
| Respiratory, thoracic and mediastinal disorders | Rhinorrhoea Rhinorrhoea Rhinorrhoea Rhinorrhoea | Nasal discharge watery excessive |
| Respiratory, thoracic and mediastinal disorders | Rhinorrhoea Chilholl | Rhinorrhea |
| Respiratory, thoracic and mediastinal disorders | Rhinorrhoea | Rhinorrhoea |
| Respiratory, thoracic and mediastinal disorders | Rhinorrhoea | Runny nose |
| Respiratory, thoracic and mediastinal disorders | Rhinorrhoea | Nasal mucus increased |
| Respiratory, thoracic and mediastinal disorders | Rhinorrhoea | Mucus nasal increased |
| Respiratory, thoracic and mediastinal disorders | Rhinorrhoea | Gustatory rhinorrhoea |
| Respiratory, thoracre and mediastinal disorders | Rhinorrhoea | Sniffles |
| Respiratory, thoracic and mediastinal disorders | Rhinorrhoea | Gustatory rhinorrhea |
| Respiratory, thoracic and mediastinal disorders | Sneezing | Paroxysmal sneeze |
| Respiratory, thoracic and mediastinal disorders | Sneezing | Sneezing |
| Respiratory, thoracic and mediastinal disorders | Sneezing | Sneezing excessive |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Respirat | ory Disorders NEC (HLT) | |
| Respiratory, thoracic and mediastinal disorders | Snoring | Snore |
| Respiratory, thoracic and mediastinal disorders | Snoring | Snoring |
| Respiratory, thoracic and mediastinal disorders | Sputum decreased | Sputum decreased |
| Respiratory, thoracic and mediastinal disorders | Sputum discoloured | Sputum discolored |
| Respiratory, thoracic and mediastinal disorders | Sputum discoloured | Sputum discoloured |
| Respiratory, thoracic and mediastinal disorders | Sputum increased | Sputum excretion increased |
| Respiratory, thoracic and mediastinal disorders | Sputum increased | Sputum increased |
| Respiratory, thoracic and mediastinal disorders | Sputum retention | Sputum excretion difficulty |
| Respiratory, thoracic and mediastinal disorders | Sputum retention Sputum retention | Sputum expectoration difficult |
| Respiratory, thoracic and mediastinal disorders | Sputum retention | Sputum sticking sensation of |
| Respiratory, thoracic and mediastinal disorders | Sputum retention | Sputum retention |
| Respiratory, thoracic and mediastinal disorders | Suffocation feeling | Suffocation feeling |
| Respiratory, thoracic and mediastinal disorders | Throat irritation | Burning in throat |
| Respiratory, thoracic and mediastinal disorders | Throat irritation | Local throat irritation |
| Respiratory, thoracic and mediastinal disorders | Throat irritation | Pharyngo-oral irritation |
| Respiratory, thoracle and mediastinal disorders | Throat irritation | Pharynx burning sensation of |
| Respiratory, thoracic and mediastinal disorders | Throat irritation | Pharynx irritated sensation of |
| Respiratory, thoracic and mediastinal disorders | Throat irritation | Pharynx itchy sensation of |
| Respiratory, thoracic and mediastinal disorders | Throat irritation | Throat burning sensation of |
| Respiratory, thoracic and mediastinal disorders | Throat irritation | Throat irritation |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Respirat | ory Disorders NEC (HLT) | |
| Respiratory, thoracic and mediastinal disorders | Throat irritation | Itchy throat |
| Respiratory, thoracic and mediastinal disorders | Throat lesion | Throat lesion |
| Respiratory, thoracic and mediastinal disorders | Throat tightness | Constriction throat |
| Respiratory, thoracic and mediastinal disorders | Throat tightness | Throat constriction |
| Respiratory, thoracic and mediastinal disorders | Throat tightness | Throat tightness |
| Respiratory, thoracic and mediastinal disorders | Upper airway necrosis | Upper airway necrosis |
| Respiratory, thoracic and mediastinal disorders | Upper airway obstruction | Upper airway obstruction |
| Respiratory, thoracic and mediastinal disorders | Upper airway resistance syndrome | Upper airway resistance syndrome |
| Respiratory, thoracic and mediastinal disorders | Upper respiratory tract congestion | Upper respiratory tract congestion |
| Respiratory, thoracic and mediastinal disorders | Upper respiratory tract inflammation | Upper respiratory tract inflammation |
| Respiratory, thoracic and mediastinal disorders | Upper respiratory tract inflammation | Acute upper respiratory tract inflammation |
| Respiratory, thoracic and mediastinal disorders | Upper respiratory tract irritation | Upper respiratory tract irritation |
| Respiratory, thoracic and mediastinal disorders | Upper-airway cough syndrome | Posterior nasal drip |
| Respiratory, thoracic and mediastinal disorders | Upper-airway cough syndrome | Postnasal drip |
| Respiratory, thoracic and mediastinal disorders | Upper-airway cough syndrome | Chronic post nasal drip |
| Respiratory, thoracic and mediastinal disorders | Upper-airway cough syndrome | Upper-airway cough syndrome |
| Respiratory, thoracic and mediastinal disorders | Yawning | Yawn |
| Respiratory, thoracic and mediastinal disorders | Yawning | Yawning |
| Respiratory, thoracic and mediastinal disorders | Yawning | Yawning excessive |

| System Organ Class | Preferred Term | Lowest Level Term |
|--------------------|----------------|-------------------|
| 15May2017 | | 63 |

| Route of Administration: Upper Respiratory Tract Disorders (HLT) (Exclude Infections) | | |
|---|---|---|
| Respiratory, thoracic and mediastinal disorders | Adductor vocal cord weakness | Adductor vocal cord weakness |
| Respiratory, thoracic and mediastinal disorders | Adenoidal disorder | Adenoidal disorder |
| Respiratory, thoracic and mediastinal disorders | Adenoidal hypertrophy | Adenoid vegetations |
| Respiratory, thoracic and mediastinal disorders | Adenoidal hypertrophy | Adenoidal hypertrophy |
| Respiratory, thoracic and mediastinal disorders | Allergic pharyngitis | Allergic pharyngitis |
| Respiratory, thoracic and mediastinal disorders | Allergic sinusitis | Allergic sinusitis |
| Respiratory, thoracic and mediastinal disorders | Allergic sinusitis | Seasonal sinusitis |
| Respiratory, thoracic and mediastinal disorders | Chronic eosinophilic rhinosinusitis | Chronic eosinophilic rhinosinusitis |
| Respiratory, thoracic and mediastinal disorders | Chronic hyperplastic eosinophilic sinusitis | Chronic hyperplastic eosinophilic sinusitis |
| Respiratory, thoracic and mediastinal disorders | Croup noninfectious | Croup noninfectious |
| Respiratory, thoracic and mediastinal disorders | Dysaesthesia pharynx | Dysaesthesia pharynx |
| Respiratory, thoracic and mediastinal disorders | Dysaesthesia pharynx | Dysesthesia pharynx |
| Respiratory, thoracic and mediastinal disorders | Dysaesthesia pharynx | Laryngopharyngeal dysesthesia |
| Respiratory, thoracic and mediastinal disorders | Dysaesthesia pharynx | Laryngopharyngeal dysaesthesia |
| Respiratory, thoracic and mediastinal disorders | Eosinophilic rhinitis | Eosinophilic rhinitis |
| Respiratory, thoracic and mediastinal disorders | Epiglottic cyst | Epiglottic cyst |
| Respiratory, thoracic and mediastinal disorders | Epiglottic erythema | Epiglottic erythema |
| Respiratory, thoracic and mediastinal disorders | Epiglottic mass | Epiglottic mass |
| Respiratory, thoracic and mediastinal disorders | Epiglottic oedema | Epiglottic oedema |
| Respiratory, thoracic and mediastinal disorders | Epiglottic oedema | Epiglottic edema |
| Respiratory, thoracic and | Epiglottis ulcer | Epiglottis ulcer |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Upper Ro | espiratory Tract Disorders (HLT) (Exc | clude Infections) |
| mediastinal disorders | | |
| Respiratory, thoracic and mediastinal disorders | Epistaxis | Bleeding nose |
| Respiratory, thoracic and mediastinal disorders | Epistaxis | Epistaxis |
| Respiratory, thoracic and mediastinal disorders | Epistaxis | Haemorrhage nasal |
| Respiratory, thoracic and mediastinal disorders | Epistaxis | Hemorrhage nasal |
| Respiratory, thoracic and mediastinal disorders | Epistaxis | Nasal bleeding |
| Respiratory, thoracic and mediastinal disorders | Epistaxis | Nasal mucus blood tinged |
| Respiratory, thoracic and mediastinal disorders | Epistaxis | Nose bleed |
| Respiratory, thoracic and mediastinal disorders | Epistaxis Epistaxis Epistaxis Epistaxis | Nose bleeds |
| Respiratory, thoracic and mediastinal disorders | Epistaxis | Nosebleed |
| Respiratory, thoracic and mediastinal disorders | Epistaxis | Chronic epistaxis |
| Respiratory, thoracic and mediastinal disorders | Intranasal hypoaesthesia | Intranasal numbness |
| Respiratory, thoracic and mediastinal disorders | Intranasal hypoaesthesia | Intranasal hypoaesthesia |
| Respiratory, thoracic and mediastinal disorders | Intranasal hypoaesthesia | Intranasal hypoesthesia |
| Respiratory, thoracic and mediastinal disorders | Intranasal paraesthesia | Intranasal paraesthesia |
| Respiratory, thoracic and mediastinal disorders | Intranasal paraesthesia | Intranasal paresthesia |
| Respiratory, thoracic and mediastinal disorders | Laryngeal cyst | Laryngeal cyst |
| Respiratory, thoracic and mediastinal disorders | Laryngeal disorder | Laryngeal disorder NOS |
| Respiratory, thoracic and mediastinal disorders | Laryngeal disorder | Unspecified disease of larynx |
| Respiratory, thoracic and mediastinal disorders | Laryngeal disorder | Laryngeal disorder |
| Respiratory, thoracic and | Laryngeal dyspnoea | Laryngeal dyspnoea |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Upper I | Respiratory Tract Disorders (HLT) (Ex | clude Infections) |
| mediastinal disorders | | |
| Respiratory, thoracic and mediastinal disorders | Laryngeal dyspnoea | Laryngeal dyspnea |
| Respiratory, thoracic and mediastinal disorders | Laryngeal erythema | Laryngeal erythema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal haematoma | Laryngeal haematoma |
| Respiratory, thoracic and mediastinal disorders | Laryngeal haematoma | Laryngeal hematoma |
| Respiratory, thoracic and mediastinal disorders | Laryngeal haematoma | Glottic haematoma |
| Respiratory, thoracic and mediastinal disorders | Laryngeal haematoma | Glottic hematoma |
| Respiratory, thoracic and mediastinal disorders | Laryngeal haemorrhage | Laryngeal haemorrhage |
| Respiratory, thoracic and mediastinal disorders | Laryngeal haemorrhage | Laryngeal hemorrhage |
| Respiratory, thoracic and mediastinal disorders | Laryngeal haemorrhage | Laryngeal bleeding |
| Respiratory, thoracic and mediastinal disorders | Laryngeal hypertrophy | Laryngeal hypertrophy |
| Respiratory, thoracic and mediastinal disorders | Laryngeal infiltration | Laryngeal infiltration NOS |
| Respiratory, thoracic and mediastinal disorders | Laryngeal infiltration | Laryngeal infiltration |
| Respiratory, thoracic and mediastinal disorders | Laryngeal inflammation | Laryngeal inflammation |
| Respiratory, thoracic and mediastinal disorders | Laryngeal inflammation | Laryngeal mucositis |
| Respiratory, thoracic and mediastinal disorders | Laryngeal leukoplakia | Laryngeal leukoplakia |
| Respiratory, thoracic and mediastinal disorders | Laryngeal leukoplakia | Laryngeal leucoplakia |
| Respiratory, thoracic and mediastinal disorders | Laryngeal mass | Laryngeal mass |
| Respiratory, thoracic and mediastinal disorders | Laryngeal necrosis | Laryngeal necrosis |
| Respiratory, thoracic and mediastinal disorders | Laryngeal necrosis | Laryngeal chondronecrosis |
| Respiratory, thoracic and | Laryngeal obstruction | Laryngeal obstruction |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Upper | Respiratory Tract Disorders (HLT) ( | (Exclude Infections) |
| mediastinal disorders | | |
| Respiratory, thoracic and mediastinal disorders | Laryngeal obstruction | Subglottic obstruction |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Edema glottis |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Edema larynx |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Edema of larynx |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Edema vocal cord |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Glottic edema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Glottic oedema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Laryngeal edema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Laryngeal oedema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Larynx edema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Larynx oedema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Oedema of larynx |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Subglottic edema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Subglottic oedema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Vocal cord edema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Vocal cord oedema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Oedema glottis |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Oedema larynx |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Oedema vocal cord |
| Respiratory, thoracic and | Laryngeal oedema | Aryepiglottis edema |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Upper l | Respiratory Tract Disorders (HLT) (E | xclude Infections) |
| mediastinal disorders | | |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Aryepiglottis oedema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Acute laryngeal edema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Acute laryngeal oedema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal polyp | Laryngeal polyp |
| Respiratory, thoracic and mediastinal disorders | Laryngeal stenosis | Laryngeal stenosis |
| Respiratory, thoracic and mediastinal disorders | Laryngeal stenosis | Laryngeal stricture |
| Respiratory, thoracic and mediastinal disorders | Laryngeal stenosis | Stenosis of larynx |
| Respiratory, thoracic and mediastinal disorders | Laryngeal stenosis | Subglottic stenosis |
| Respiratory, thoracic and mediastinal disorders | Laryngeal stenosis | Supraglottic stenosis |
| Respiratory, thoracic and mediastinal disorders | Laryngeal ulceration | Laryngeal ulceration |
| Respiratory, thoracic and mediastinal disorders | Laryngeal ulceration | Larynx ulcer |
| Respiratory, thoracic and mediastinal disorders | Laryngeal ulceration | Larynx ulceration |
| Respiratory, thoracic and mediastinal disorders | Laryngeal ventricle prolapse | Laryngeal ventricle prolapse |
| Respiratory, thoracic and mediastinal disorders | Laryngitis allergic | Laryngitis allergic |
| Respiratory, thoracic and mediastinal disorders | Laryngospasm | Glottic spasm |
| Respiratory, thoracic and mediastinal disorders | Laryngospasm | Laryngeal spasm |
| Respiratory, thoracic and mediastinal disorders | Laryngospasm | Laryngismus |
| Respiratory, thoracic and mediastinal disorders | Laryngospasm | Laryngospasm |
| Respiratory, thoracic and mediastinal disorders | Laryngospasm | Larynx muscle hypersensitive |
| Respiratory, thoracic and | Laryngospasm | Spasm glottis |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Upper | Respiratory Tract Disorders (HLT) | (Exclude Infections) |
| mediastinal disorders | | |
| Respiratory, thoracic and mediastinal disorders | Laryngospasm | Spasm larynx |
| Respiratory, thoracic and mediastinal disorders | Larynx irritation | Larynx irritation |
| Respiratory, thoracic and mediastinal disorders | Larynx irritation | Larynx itching |
| Respiratory, thoracic and mediastinal disorders | Maxillary sinus pseudocyst | Maxillary sinus pseudocyst |
| Respiratory, thoracic and mediastinal disorders | Nasal cavity mass | Nasal cavity mass |
| Respiratory, thoracic and mediastinal disorders | Nasal congestion | Congestion nasal |
| Respiratory, thoracic and mediastinal disorders | Nasal congestion | Nasal congestion |
| Respiratory, thoracic and mediastinal disorders | Nasal congestion | Nasal stuffiness |
| Respiratory, thoracic and mediastinal disorders | Nasal congestion Nasal congestion | Nose congestion |
| Respiratory, thoracic and mediastinal disorders | Nasal congestion | Rhinitis medicamentosa |
| Respiratory, thoracic and mediastinal disorders | Nasal congestion | Rhinitis medicamentous |
| Respiratory, thoracic and mediastinal disorders | Nasal congestion | Nasal mucosal swelling |
| Respiratory, thoracic and mediastinal disorders | Nasal congestion | Chronic nasal congestion |
| Respiratory, thoracic and mediastinal disorders | Nasal congestion | Acute nasal congestion |
| Respiratory, thoracic and mediastinal disorders | Nasal cyst | Nasal cyst |
| Respiratory, thoracic and mediastinal disorders | Nasal cyst | Intranasal cyst |
| Respiratory, thoracic and mediastinal disorders | Nasal disorder | Nasal disorder NOS |
| Respiratory, thoracic and mediastinal disorders | Nasal disorder | Nasal disorder |
| Respiratory, thoracic and mediastinal disorders | Nasal dryness | Dry nose |
| Respiratory, thoracic and | Nasal dryness | Nasal dryness |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Upper | Respiratory Tract Disorders (HLT) (Ex | clude Infections) |
| mediastinal disorders | | |
| Respiratory, thoracic and mediastinal disorders | Nasal dryness | Nose dry feeling of |
| Respiratory, thoracic and mediastinal disorders | Nasal dryness | Nose dryness |
| Respiratory, thoracic and mediastinal disorders | Nasal inflammation | Nasal inflammation |
| Respiratory, thoracic and mediastinal disorders | Nasal inflammation | Nasal septal inflammation |
| Respiratory, thoracic and mediastinal disorders | Nasal inflammation | Nasal mucosal inflammation |
| Respiratory, thoracic and mediastinal disorders | Nasal mucosa atrophy | Nasal mucosa atrophy |
| Respiratory, thoracic and mediastinal disorders | Nasal mucosal discolouration | Nasal mucosal discolouration |
| Respiratory, thoracic and mediastinal disorders | Nasal mucosal discolouration | Nasal mucosal discoloration |
| Respiratory, thoracic and mediastinal disorders | Nasal mucosal discolouration | Nasal mucosal pallor |
| Respiratory, thoracic and mediastinal disorders | Nasal mucosal disorder | Nasal mucosal disorder NOS |
| Respiratory, thoracic and mediastinal disorders | Nasal mucosal disorder | Nasal mucosal disorder |
| Respiratory, thoracic and mediastinal disorders | Nasal mucosal disorder | Nasal mucosal erythema |
| Respiratory, thoracic and mediastinal disorders | Nasal mucosal disorder | Nasal mucosal hyperaemia |
| Respiratory, thoracic and mediastinal disorders | Nasal mucosal disorder | Nasal mucosal ulcer |
| Respiratory, thoracic and mediastinal disorders | Nasal mucosal disorder | Nasal mucosal hyperemia |
| Respiratory, thoracic and mediastinal disorders | Nasal mucosal hypertrophy | Nasal mucosal hypertrophy |
| Respiratory, thoracic and mediastinal disorders | Nasal necrosis | Nasal mucosal necrosis |
| Respiratory, thoracic and mediastinal disorders | Nasal necrosis | Nasal necrosis |
| Respiratory, thoracic and mediastinal disorders | Nasal necrosis | Necrosis nasal |
| Respiratory, thoracic and | Nasal necrosis | Nasal septal mucosa necrosis |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Upper Respiratory Tract Disorders (HLT) (Exclude Infections) | | |
| mediastinal disorders | | |
| Respiratory, thoracic and mediastinal disorders | Nasal odour | Nasal odour |
| Respiratory, thoracic and mediastinal disorders | Nasal odour | Nasal odor |
| Respiratory, thoracic and mediastinal disorders | Nasal oedema | Nasal oedema |
| Respiratory, thoracic and mediastinal disorders | Nasal oedema | Nose edema |
| Respiratory, thoracic and mediastinal disorders | Nasal oedema | Nose oedema |
| Respiratory, thoracic and mediastinal disorders | Nasal oedema | Nasal turbinate edema |
| Respiratory, thoracic and mediastinal disorders | Nasal oedema | Nasal edema |
| Respiratory, thoracic and mediastinal disorders | Nasal oedema Nasal polyps Nasal polyps | Nasal turbinate oedema |
| Respiratory, thoracic and mediastinal disorders | Nasal polyps | Nasal polyp |
| Respiratory, thoracic and mediastinal disorders | Nasal polyps | Nasal polyps |
| Respiratory, thoracic and mediastinal disorders | Nasal polyps | Polyp of nasal cavity |
| Respiratory, thoracic and mediastinal disorders | Nasal polyps | Polyps nasal |
| Respiratory, thoracic and mediastinal disorders | Nasal polyps | Unspecified nasal polyp |
| Respiratory, thoracic and mediastinal disorders | Nasal polyps | Hyperplastic nasal polyp |
| Respiratory, thoracic and mediastinal disorders | Nasal polyps | Choanal polyp |
| Respiratory, thoracic and mediastinal disorders | Nasal septum disorder | Nasal septum disorder |
| Respiratory, thoracic and mediastinal disorders | Nasal septum disorder | Nasal septum disorder NOS |
| Respiratory, thoracic and mediastinal disorders | Nasal septum disorder | Nasal septal erythema |
| Respiratory, thoracic and mediastinal disorders | Nasal septum perforation | Nasal septum perforation |
| Respiratory, thoracic and | Nasal septum perforation | Perforation nasal septum |

| System Organ Class | Preferred Term | Lowest Level Term | | |
|---|---|---|--|--|
| Route of Administration: Upper Respiratory Tract Disorders (HLT) (Exclude Infections) | | | | |
| mediastinal disorders | | | | |
| Respiratory, thoracic and mediastinal disorders | Nasal septum ulceration | Nasal septum ulceration | | |
| Respiratory, thoracic and mediastinal disorders | Nasal turbinate abnormality | Nasal turbinate abnormality | | |
| Respiratory, thoracic and mediastinal disorders | Nasal turbinate hypertrophy | Hypertrophy of nasal turbinates | | |
| Respiratory, thoracic and mediastinal disorders | Nasal turbinate hypertrophy | Nasal turbinate hypertrophy | | |
| Respiratory, thoracic and mediastinal disorders | Nasal turbinate hypertrophy | Concha bullosa | | |
| Respiratory, thoracic and mediastinal disorders | Nasal ulcer | Nasal ulcer | | |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal spasm | Oropharyngeal spasm | | |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal spasm | Spasm oropharyngeal | | |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal swelling | Oropharyngeal swelling | | |
| Respiratory, thoracic and mediastinal disorders | Paranasal cyst | Paranasal sinus mucocoele | | |
| Respiratory, thoracic and mediastinal disorders | Paranasal cyst | Paranasal cyst | | |
| Respiratory, thoracic and mediastinal disorders | Paranasal cyst | Paranasal sinus mucocele | | |
| Respiratory, thoracic and mediastinal disorders | Paranasal sinus haematoma | Maxillary sinus haematoma | | |
| Respiratory, thoracic and mediastinal disorders | Paranasal sinus haematoma | Maxillary sinus hematoma | | |
| Respiratory, thoracic and mediastinal disorders | Paranasal sinus haematoma | Paranasal sinus haematoma | | |
| Respiratory, thoracic and mediastinal disorders | Paranasal sinus haematoma | Paranasal sinus hematoma | | |
| Respiratory, thoracic and mediastinal disorders | Paranasal sinus hypersecretion | Paranasal sinus hypersecretion | | |
| Respiratory, thoracic and mediastinal disorders | Paranasal sinus hypersecretion | Nasal sinus discharge | | |
| Respiratory, thoracic and mediastinal disorders | Paranasal sinus mucosal hypertrophy | Paranasal sinus mucosal hypertrophy | | |
| Respiratory, thoracic and | Paranasal sinus necrosis | Paranasal sinus necrosis | | |
| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Upper | Respiratory Tract Disorders (HLT) (Ex | xclude Infections) |
| mediastinal disorders | | |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal cyst | Pharyngeal cyst |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal disorder | Pharyngeal disorder NOS |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal disorder | Unspecified disease of pharynx |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal disorder | Nasopharyngeal disorder |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal disorder | Pharyngeal disorder |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal dyskinesia | Pharyngeal dyskinesia |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal enanthema | Pharyngeal enanthema |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal erosion | Pharyngeal erosion |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal erythema | Pharynx redness of |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal crythema | Red throat |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal crythema | Pharyngeal erythema |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal erythema | Uvular erythema |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal exudate | Pharyngeal exudate |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal fistula | Pharyngeal fistula |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal haematoma | Pharyngeal haematoma |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal haematoma | Pharyngeal hematoma |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal haemorrhage | Haemorrhage from throat |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal haemorrhage | Haemorrhage pharyngeal |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal haemorrhage | Hemorrhage from throat |
| Respiratory, thoracic and | Pharyngeal haemorrhage | Pharyngeal haemorrhage |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Upper | Respiratory Tract Disorders (HLT) (Ex | clude Infections) |
| mediastinal disorders | | |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal haemorrhage | Hemorrhage pharyngeal |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal haemorrhage | Pharyngeal hemorrhage |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal haemorrhage | Oropharyngeal hemorrhage |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal haemorrhage | Oropharyngeal haemorrhage |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal haemorrhage | Pharyngeal bleeding |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal hypertrophy | Pharyngeal hypertrophy |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal hypoaesthesia | Pharyngeal hypoaesthesia |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal hypoaesthesia | Numbness throat |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal hypoaesthesia | Pharyngeal hypoesthesia |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal inflammation | Pharyngeal inflammation |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal inflammation | Pharyngeal mucositis |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal lesion | Pharyngeal lesion |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal leukoplakia | Pharyngeal leukoplakia |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal mass | Pharyngeal mass |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal mucosa atrophy | Pharyngeal mucosa atrophy |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal necrosis | Pharyngeal necrosis |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal oedema | Edema pharynx |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal oedema | Oedema pharynx |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal oedema | Pharyngeal oedema |
| Respiratory, thoracic and | Pharyngeal oedema | Pharynx edema |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Upper l | Respiratory Tract Disorders (HLT) (E | Exclude Infections) |
| mediastinal disorders | | |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal oedema | Throat edema |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal oedema | Throat oedema |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal oedema | Throat swelling |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal oedema | Throat swelling non-specific |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal oedema | Throat swelling NOS |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal oedema | Pharyngeal edema |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal oedema | Pharynx oedema |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal polyp | Pharyngeal polyp |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal stenosis | Pharyngeal stenosis |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal decration | Pharyngeal ulceration |
| Respiratory, thoracic and mediastinal disorders | Reflux laryngitis | Laryngopharyngeal reflux |
| Respiratory, thoracic and mediastinal disorders | Reflux laryngitis | Reflux laryngitis |
| Respiratory, thoracic and mediastinal disorders | Rhinitis allergic | Allergic rhinitis |
| Respiratory, thoracic and mediastinal disorders | Rhinitis allergic | Allergic rhinitis (excl hay fever) |
| Respiratory, thoracic and mediastinal disorders | Rhinitis allergic | Atopic rhinitis |
| Respiratory, thoracic and mediastinal disorders | Rhinitis allergic | Rhinitis allergic |
| Respiratory, thoracic and mediastinal disorders | Rhinitis allergic | Rhinitis allergic atopic |
| Respiratory, thoracic and mediastinal disorders | Rhinitis allergic | Rhinitis allergic NOS |
| Respiratory, thoracic and mediastinal disorders | Rhinitis atrophic | Atrophic rhinitis |
| Respiratory, thoracic and | Rhinitis atrophic | Ozena |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Upper | Respiratory Tract Disorders (HLT) | (Exclude Infections) |
| mediastinal disorders | | |
| Respiratory, thoracic and mediastinal disorders | Rhinitis atrophic | Rhinitis atrophic |
| Respiratory, thoracic and mediastinal disorders | Rhinitis atrophic | Dry rhinitis |
| Respiratory, thoracic and mediastinal disorders | Rhinitis hypertrophic | Rhinitis hypertrophic |
| Respiratory, thoracic and mediastinal disorders | Rhinitis perennial | Perennial allergic rhinitis |
| Respiratory, thoracic and mediastinal disorders | Rhinitis perennial | Perennial rhinitis |
| Respiratory, thoracic and mediastinal disorders | Rhinitis perennial | Rhinitis perennial |
| Respiratory, thoracic and mediastinal disorders | Rhinitis seasonal | Allergic rhinitis due to pollen |
| Respiratory, thoracic and mediastinal disorders | Rhinitis seasonal | Rhinitis seasonal |
| Respiratory, thoracic and mediastinal disorders | Rhinitis seasonal | Seasonal allergic rhinitis |
| Respiratory, thoracic and mediastinal disorders | Rhinitis seasonal | Seasonal rhinitis |
| Respiratory, thoracic and mediastinal disorders | Rhinitis ulcerative | Rhinitis ulcerative |
| Respiratory, thoracic and mediastinal disorders | Rhinolithiasis | Rhinolithiasis |
| Respiratory, thoracic and mediastinal disorders | Rhinolithiasis | Nasal calculus |
| Respiratory, thoracic and mediastinal disorders | Sinus congestion | Nasal sinus congestion |
| Respiratory, thoracic and mediastinal disorders | Sinus congestion | Sinus congestion |
| Respiratory, thoracic and mediastinal disorders | Sinus disorder | Sinus disorder NOS |
| Respiratory, thoracic and mediastinal disorders | Sinus disorder | Sinus disorder |
| Respiratory, thoracic and mediastinal disorders | Sinus perforation | Perforation of sinus |
| Respiratory, thoracic and mediastinal disorders | Sinus perforation | Sinus perforation |
| Respiratory, thoracic and | Sinus polyp | Antral polyp (of maxillary sinus) |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Upper | Respiratory Tract Disorders (HLT) ( | (Exclude Infections) |
| mediastinal disorders | | |
| Respiratory, thoracic and mediastinal disorders | Sinus polyp | Maxillary sinus polyp |
| Respiratory, thoracic and mediastinal disorders | Sinus polyp | Sinus polyp |
| Respiratory, thoracic and mediastinal disorders | Sinus polyp degeneration | Polypoid sinus degeneration |
| Respiratory, thoracic and mediastinal disorders | Sinus polyp degeneration | Sinus polyp degeneration |
| Respiratory, thoracic and mediastinal disorders | Sinusitis noninfective | Sinusitis noninfective |
| Respiratory, thoracic and mediastinal disorders | Stridor | Stridor |
| Respiratory, thoracic and mediastinal disorders | Stridor | Stridor inspiratory |
| Respiratory, thoracic and mediastinal disorders | Tonsillar atrophy | Tonsillar atrophy |
| Respiratory, thoracic and mediastinal disorders | Tonsillar atrophy | Submerged tonsil |
| Respiratory, thoracic and mediastinal disorders | Tonsillar disorder | Chronic tonsillar disease |
| Respiratory, thoracic and mediastinal disorders | Tonsillar disorder | Tonsillar disorder |
| Respiratory, thoracic and mediastinal disorders | Tonsillar disorder | Cryptic tonsil |
| Respiratory, thoracic and mediastinal disorders | Tonsillar haemorrhage | Tonsillar haemorrhage |
| Respiratory, thoracic and mediastinal disorders | Tonsillar haemorrhage | Tonsillar hemorrhage |
| Respiratory, thoracic and mediastinal disorders | Tonsillar haemorrhage | Tonsillar bleeding |
| Respiratory, thoracic and mediastinal disorders | Tonsillar hypertrophy | Tonsillar hypertrophy |
| Respiratory, thoracic and mediastinal disorders | Tonsillar hypertrophy | Enlarged tonsils |
| Respiratory, thoracic and mediastinal disorders | Tonsillar inflammation | Tonsillar inflammation |
| Respiratory, thoracic and mediastinal disorders | Tonsillar ulcer | Tonsillar ulcer |
| Respiratory, thoracic and | Tonsillolith | Tonsillolith |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Upper | Respiratory Tract Disorders (HLT) ( | <b>Exclude Infections)</b> |
| mediastinal disorders | | |
| Respiratory, thoracic and mediastinal disorders | Vasomotor rhinitis | Vasomotor rhinitis |
| Respiratory, thoracic and mediastinal disorders | Velopharyngeal incompetence | Velopharyngeal incompetence |
| Respiratory, thoracic and mediastinal disorders | Vocal cord atrophy | Vocal cord atrophy |
| Respiratory, thoracic and mediastinal disorders | Vocal cord cyst | Vocal cord cyst |
| Respiratory, thoracic and mediastinal disorders | Vocal cord disorder | Vocal cord disorder NOS |
| Respiratory, thoracic and mediastinal disorders | Vocal cord disorder | Vocal cord dysfunction |
| Respiratory, thoracic and mediastinal disorders | Vocal cord disorder | Vocal cord disorder |
| Respiratory, thoracic and mediastinal disorders | Vocal cord inflammation | Vocal cord inflammation |
| Respiratory, thoracic and mediastinal disorders | Vocal cord leukoplakia | Vocal cord leukoplakia |
| Respiratory, thoracic and mediastinal disorders | Vocal cord polyp | Polyp of vocal cord |
| Respiratory, thoracic and mediastinal disorders | Vocal cord polyp | Vocal cord polyp |
| Respiratory, thoracic and mediastinal disorders | Vocal cord thickening | Singers nodules |
| Respiratory, thoracic and mediastinal disorders | Vocal cord thickening | Vocal cord thickening |
| Respiratory, thoracic and mediastinal disorders | Vocal cord thickening | Vocal cord nodule |

## (4) AEs related to taste and smell disorders:

| System Organ Class | Preferred Term | Lowest Level Term |
|---------------------------------|----------------|-------------------------|
| Taste and Smell Disorders (SMQ) | | |
| Nervous system disorders | Dysgeusia | After taste |
| Nervous system disorders | Ageusia | Ageusia |
| Nervous system disorders | Parosmia | Altered smell sensation |
| Nervous system disorders | Anosmia | Anosmia |
| Nervous system disorders | Dysgeusia | Dysgeusia |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Taste and Smell Disorders (SMQ) | | |
| Nervous system disorders | Parosmia | Dysosmia |
| Nervous system disorders | Parosmia | Dysosmia NOS |
| Nervous system disorders | Parosmia | Faint odor of sulfur |
| Nervous system disorders | Hypogeusia | Gustatory sense diminished |
| Psychiatric disorders | Hallucination, gustatory | Hallucination gustatory |
| Psychiatric disorders | Hallucination, olfactory | Hallucination olfactory |
| Psychiatric disorders | Hallucination, gustatory | Hallucination, gustatory |
| Psychiatric disorders | Hallucination, olfactory | Hallucination, olfactory |
| Nervous system disorders | Parosmia | Hyperosmia |
| Nervous system disorders | Hypogeusia | Hypogeusia |
| Nervous system disorders | Anosmia | Loss of smell |
| Nervous system disorders | Ageusia | Loss of taste |
| Psychiatric disorders | Hallucination, olfactory | Olfactory hallucination |
| Nervous system disorders | Hallucination, olfactory Dysgeusia Parosmia Parosmia Parosmia Parosmia | Parageusia |
| Nervous system disorders | Parosmia | Parosmia |
| Nervous system disorders | Parosmia C MO | Perversion olfactory |
| Nervous system disorders | Parosmia | Smell alteration |
| Nervous system disorders | Parosmia | Smell change |
| Nervous system disorders | Anosmia | Smell loss |
| Nervous system disorders | Parosmia | Smell perversion |
| Nervous system disorders | Parosmia | Smelly sensation |
| Nervous system disorders | Parosmia | Strange smell sensation |
| Nervous system disorders | Dysgeusia | Taste abnormality |
| Nervous system disorders | Ageusia | Taste absent |
| Nervous system disorders | Dysgeusia | Taste alteration |
| Nervous system disorders | Dysgeusia | Taste altered |
| Nervous system disorders | Dysgeusia | Taste bitter |
| Nervous system disorders | Dysgeusia | Taste bitter-salty |
| Nervous system disorders | Dysgeusia | Taste changed |
| Nervous system disorders | Hypogeusia | Taste diminished |
| Nervous system disorders | Dysgeusia | Taste disturbance |
| Nervous system disorders | Dysgeusia | Taste garlic |
| Nervous system disorders | Ageusia | Taste loss |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Taste and Smell Disorders (SMQ) | | |
| Nervous system disorders | Dysgeusia | Taste metallic |
| Nervous system disorders | Dysgeusia | Taste peculiar |
| Nervous system disorders | Dysgeusia | Taste perversion |
| Nervous system disorders | Dysgeusia | Taste salty |
| Nervous system disorders | Dysgeusia | Taste sour |
| Nervous system disorders | Dysgeusia | Taste sweet |
| Nervous system disorders | Dysgeusia | Bilious taste |
| Nervous system disorders | Parosmia | Cacosmia |
| Nervous system disorders | Hyposmia | Hyposmia |
| Nervous system disorders | Parosmia | Faint odour of sulfur |
| Nervous system disorders | Olfactory nerve disorder | Olfactory nerve disorder |
| Investigations | Olfactory test abnormal | Olfactory test abnormal |
| Investigations | Olfactory test abnormal | Olfactory acuity test abnormal |
| Nervous system disorders | Hyposmia | Diminished sense of smell |
| Investigations | Olfactory test abnormal Hyposmia Gustometry abnormal | Gustometry abnormal |
| General disorders and administration site conditions | Product taste abnormat | Medication after taste |
| Nervous system disorders | Parosmia | Phantosmia |
| Nervous system disorders | Parosmia | Olfactism |
| Nervous system disorders | Hypergeusia | Hypergeusia |
| Nervous system disorders | Dysgeusia | Chalky taste |

(5) AEs related to depression and suicidality/self-injury:

| Preferred Term | Lowest Level Term |
|---|---|
| Depression and Suicide/Self-Injury: Depression (SMQ) (Exclude Suicide/Self-Injury) | |
| Activation syndrome | Activation syndrome |
| Adjustment disorder with depressed mood | Adjustment disorder with depressed mood |
| Adjustment disorder with depressed mood | Adjustment reaction with brief depressive reaction |
| Adjustment disorder with depressed mood | Adjustment reaction with prolonged depressive reaction |
| Adjustment disorder with mixed anxiety and depressed mood | Adjustment disorder with mixed anxiety and depressed mood |
| Agitated depression | Agitated depression |
| Agitated depression | Depression agitated |
| Anhedonia | Anhedonia |

15May2017 80

| Preferred Term | Lowest Level Term |
|---|---|
| Depression and Suicide/Self-Injury: Depression (SMQ | ) (Exclude Suicide/Self-Injury) |
| Anhedonia | Loss of all pleasure |
| Antidepressant therapy | Antidepressant therapy |
| Childhood depression | Childhood depression |
| Decreased interest | Decreased interest |
| Decreased interest | Loss of all interest |
| Decreased interest | Loss of interest |
| Decreased interest | Reduced interest in usual activities |
| Depressed mood | Chronic depressive mood |
| Depressed mood | Dejection emotional |
| Depressed mood | Depressed mood |
| Depressed mood | Emotional dejection |
| Depressed mood | Feeling blue |
| Depressed mood | Feeling down |
| Depressed mood | Feeling sad |
| Depressed mood | Low mood |
| Depressed mood | Mood depression |
| Depressed mood | Mood depressions |
| Depressed mood | Unhappiness |
| Depression | Acute depression |
| Depression | Anxiety depression |
| Depression | Anxiodepressive syndrome |
| Depression | Anxious depression |
| Depression | Atypical depressive disorder |
| Depression | Brief depressive reaction |
| Depression | Chronic depression |
| Depression | Depressed reaction |
| Depression | Depressed state |
| Depression | Depression |
| Depression | Depression aggravated |
| Depression | Depression functional |
| Depression | Depression mental |
| Depression | Depression NOS |
| Depression | Depression reactive |

15May2017

| Preferred Term | Lowest Level Term |
|---|---|
| Depression and Suicide/Self-Injury: Depression (SMC | 2) (Exclude Suicide/Self-Injury) |
| Depression | Depression worsened |
| Depression | Depressive disorder |
| Depression | Depressive episode |
| Depression | Depressive illness |
| Depression | Depressive reaction |
| Depression | Depressive state |
| Depression | Depressive stupor |
| Depression | Exogenous depression |
| Depression | Mixed anxiety & depressive |
| Depression | Reactive depression |
| Depression | Recurrent depressive disorder |
| Depression | Unipolar depression |
| Depression | Unipolar depressive illness |
| Depression postoperative | Depression postoperative |
| Depression postoperative | Postoperative depression |
| Depressive symptoms | Depressive symptoms |
| Depressive symptoms | Depressive symptoms aggravvated |
| Dysphoria | Dysphoria |
| Dysthymic disorder | Chronic depressive personality disorder |
| Dysthymic disorder | Depression neurotic |
| Dysthymic disorder | Depressive neurosis |
| Dysthymic disorder | Depressive personality disorder |
| Dysthymic disorder | Dysthymia |
| Dysthymic disorder | Dysthymic disorder |
| Dysthymic disorder | Neurotic depression |
| Electroconvulsive therapy | Bilateral ECT |
| Electroconvulsive therapy | ECT |
| Electroconvulsive therapy | ECT (electro-convulsive therapy) |
| Electroconvulsive therapy | Electroconvulsive therapy |
| Electroconvulsive therapy | Modified ECT |
| Electroconvulsive therapy | Unilateral ECT |
| Electroconvulsive therapy | Unmodified ECT |
| Feeling guilty | Feeling guilty |

| Preferred Term | Lowest Level Term |
|---|---|
| Depression and Suicide/Self-Injury: Depression (SI | MQ) (Exclude Suicide/Self-Injury) |
| Feeling guilty | Feeling remorse |
| Feeling of despair | Feeling of despair |
| Feelings of worthlessness | Feelings of worthlessness |
| Major depression | Depression endogenous |
| Major depression | Depression psychotic |
| Major depression | Depressive type psychosis |
| Major depression | Endogenous depression |
| Major depression | Involutional depression |
| Major depression | Involutional melancholia |
| Major depression | Major depression |
| Major depression | Major depressive disorder aggravated |
| Major depression | Major depressive disorder NOS |
| Major depression | Major depressive disorder with melancholic features |
| Major depression | Major depressive disorder, recurrent episode |
| Major depression | Major depressive disorder, recurrent episode, in full remission |
| Major depression | Major depressive disorder, single episode |
| Major depression Major depression Major depression | Major depressive disorder, single episode in full remission |
| Major depression | Major depressive illness |
| Major depression | Melancholia |
| Major depression | Melancholic depression |
| Major depression | Psychosis depressive |
| Major depression | Psychotic depression |
| Menopausal depression | Depression perimenopausal |
| Menopausal depression | Depression postmenopausal |
| Menopausal depression | Menopausal depression |
| Menopausal depression | Postmenopausal depression |
| Post stroke depression | Post stroke depression |
| Postictal depression | Postictal depression |
| Postpartum depression | Baby blues |
| Postpartum depression | Depression puerperal |
| Postpartum depression | Postnatal blues |
| Postpartum depression | Postnatal depression (excl psychosis) |
| 15May2017 | 83 |

| Preferred Term | Lowest Level Term |
|---|---|
| Depression and Suicide/Self-Injury: Depression (S | MQ) (Exclude Suicide/Self-Injury) |
| Postpartum depression | Postpartum depression |
| Postpartum depression | Puerperal depression |
| Postpartum depression | Transitory postpartum mood disturbance |
| Affect lability | Affect lability |
| Affect lability | Affective incontinence |
| Affect lability | Emotional incontinence |
| Affect lability | Emotional instability |
| Affect lability | Emotional lability |
| Affect lability | Instability emotional |
| Affect lability | Labile affect |
| Affect lability | Lability emotional |
| Affect lability | Mental lability symptom |
| Affect lability | Pseudobulbar affect |
| Alcohol abuse | Alcohol abuse |
| Alcohol abuse | Alcohol abuse chronic |
| Alcohol abuse | Atcohol abuse, continuous drinking behavior |
| Alcohol abuse | Alcohol abuse, continuous drinking behaviour |
| Alcohol abuse | Alcohol abuse, episodic drinking behavior |
| Alcohol abuse | Alcohol abuse, episodic drinking behaviour |
| Alcohol abuse | Alcohol abuse, in remission |
| Alcohol abuse | Alcohol abuse, unspecified drinking behavior |
| Alcohol abuse | Alcohol abuse, unspecified drinking behaviour |
| Alcohol abuse | Nondependent abuse of alcohol |
| Alcohol poisoning | Acute alcoholic intoxication |
| Alcohol poisoning | Acute alcoholic intoxication in alcoholism, continuous drinking behavior |
| Alcohol poisoning | Acute alcoholic intoxication in alcoholism, continuous drinking behaviour |
| Alcohol poisoning | Acute alcoholic intoxication in alcoholism, episodic drinking behavior |
| Alcohol poisoning | Acute alcoholic intoxication in alcoholism, episodic drinking behaviour |
| Alcohol poisoning | Acute alcoholic intoxication in alcoholism, in remission |
| Alcohol poisoning | Acute alcoholic intoxication in alcoholism, unspecified drinking behavior |
| 15May2017 | 84 |

| Preferred Term | Lowest Level Term |
|---|---|
| Depression and Suicide/Self-Injury: Depression (SMC | Q) (Exclude Suicide/Self-Injury) |
| Alcohol poisoning | Acute alcoholic intoxication in alcoholism, unspecified drinking behaviour |
| Alcohol poisoning | Alcohol intoxication |
| Alcohol poisoning | Alcohol intoxication acute |
| Alcohol poisoning | Alcohol intoxication, acute |
| Alcohol poisoning | Alcohol poisoning |
| Alcohol poisoning | Drunkenness |
| Alcohol poisoning | Toxic effect of alcohol |
| Alcohol poisoning | Toxic effect of ethyl alcohol |
| Alcohol poisoning | Toxic effect of fusel oil |
| Alcohol poisoning | Toxic effect of isopropyl alcohol |
| Alcohol poisoning | Toxic effect of methyl alcohol |
| Alcohol poisoning | Toxic effect of unspecified alcohol |
| Alcohol problem | Alcohol problem |
| Alcohol problem | Alcohol problem NOS |
| Alcohol rehabilitation | Alcohol rehabilitation |
| Alcoholism | Alcohol addiction |
| Alcoholism | Alcohol craving |
| Alcoholism | Alcohol dependence syndrome |
| Alcoholism | Alcoholic relapse |
| Alcoholism | Alcoholism |
| Alcoholism | Alcoholism (excl psychosis) |
| Alcoholism | Chronic alcoholism |
| Alcoholism | Dipsomania |
| Apathy | Ambition loss of |
| Apathy | Apathy |
| Apathy Clot | Avolition |
| Apathy Co | Initiative loss of |
| Apathy | Lack of motivation |
| Apathy | Loss of ambition |
| Apathy | Loss of initiative |
| Blunted affect | Affective blunting |
| Blunted affect | Blunted affect |

| Preferred Term | Lowest Level Term |
|---|---|
| Depression and Suicide/Self-Injury: Depression ( | SMQ) (Exclude Suicide/Self-Injury) |
| Constricted affect | Constricted affect |
| Constricted affect | Restricted affect |
| Crying | Crying |
| Crying | Crying abnormal |
| Crying | Crying uncontrollable |
| Crying | High-pitched crying |
| Crying | Inconsolable crying |
| Crying | Persistent crying |
| Crying | Uncontrollable crying |
| Crying | Weeping |
| Crying | Weepy |
| Disturbance in attention | Attention concentration difficulty |
| Disturbance in attention | Attention impaired |
| Disturbance in attention | Attentiveness decreased |
| Disturbance in attention | Concentration (mental) abnormal |
| Disturbance in attention | Concentration ability impaired |
| Disturbance in attention | Concentration impaired |
| Disturbance in attention | Concentration impairment |
| Disturbance in attention | Concentration loss |
| Disturbance in attention | Disturbance in attention |
| Disturbance in attention | Impairment of attention |
| Disturbance in attention | Mental concentration decreased |
| Disturbance in attention | Mental concentration difficult |
| Disturbance in attention | Mental concentration difficulty |
| Disturbance in attention | Mental concentration impaired |
| Disturbance in attention | Poor concentration |
| Disturbance in attention | Simple disturbance of activity and attention |
| Disturbance in attention | Vigilance decreased |
| Dyssomnia | Dysfunctions associated with sleep stages or arousal from sleep |
| Dyssomnia | Dyssomnia |
| Dyssomnia | Dyssomnia NOS |
| Emotional distress | Embarrassment |
| | 1 |

| Preferred Term | Lowest Level Term |
|---|---|
| Depression and Suicide/Self-Injury: Depression (SMC | (2) (Exclude Suicide/Self-Injury) |
| Emotional distress | Emotional distress |
| Emotional distress | Humiliation |
| Emotional distress | Mental distress |
| Emotional distress | Suffering |
| Emotional poverty | Emotional poverty |
| Emotional poverty | Emotional withdrawal |
| Emotional poverty | Lack of feeling emotions |
| Emotional poverty | Poverty emotional |
| Emotional poverty | Withdrawal emotional |
| Hypersomnia | Hypersomnia |
| Hypersomnia | Idiopathic hypersomnia |
| Hypersomnia | Persistent disorder of initiating or maintaining wakefulness |
| Hypersomnia | Primary hypersomnia |
| Hypersomnia | Sleep excessive |
| Hypersomnia | Transient disorder of initiating or maintaining wakefulness |
| Hyposomnia Impaired self-care Initial insomnia Initial insomnia | Hyposomnia |
| Impaired self-care | Impaired self-care |
| Initial insomnia | Initial insomnia |
| Initial insomnia | Trouble falling asleep |
| Intentional product misuse | Intentional drug misuse |
| Intentional product misuse | Intentional misuse |
| Intentional product misuse | Intentional misuse by dose change |
| Intentional product misuse | Intentional misuse in dosing frequency |
| Intentional product misuse | Intentional product misuse |
| Intentional product use issue | Intentional dose decrease |
| Intentional product use issue | Intentional dose increase |
| Intentional product use issue | Intentional product use issue |
| Intentional product use issue | Intentional use beyond labeled administration duration |
| Intentional product use issue | Intentional use beyond labeled duration |
| Intentional product use issue | Intentional use beyond labelled administration duration |
| Intentional product use issue | Intentional use beyond labelled duration |
| Intentional product use issue | Intentional use by incorrect route |
| 15May2017 | 87 |

| Preferred Term | Lowest Level Term |
|---|---|
| Depression and Suicide/Self-Injury: Depression (SMQ | ) (Exclude Suicide/Self-Injury) |
| Intentional product use issue | Intentional use for unlabeled indication |
| Intentional product use issue | Intentional use for unlabelled indication |
| Listless | Listless |
| Listless | Listlessness |
| Maternal use of illicit drugs | Maternal use of illicit drugs |
| Memory impairment | Forgetfulness |
| Memory impairment | Hypomnesia |
| Memory impairment | Memory deficit |
| Memory impairment | Memory disturbance |
| Memory impairment | Memory disturbance (excl dementia) |
| Memory impairment | Memory impaired |
| Memory impairment | Memory impairment |
| Memory impairment | Short-term memory impairment |
| Middle insomnia | Arousal night |
| Middle insomnia | Middle insomnia |
| Middle insomnia | Nocturnal awakening |
| Middle insomnia | Sleep maintenance insomnia |
| Mood altered | Affect alteration |
| Mood altered | Affect altered |
| Mood altered | Altered mood |
| Mood altered | Bad mood |
| Mood altered | Mood alteration NOS |
| Mood altered | Mood altered |
| Mood altered | Mood change |
| Mood swings | Mood swings |
| Mood swings | Mood variable |
| Morose and | Morose |
| Morose | Moroseness |
| Negative thoughts | Negative thoughts |
| Neglect of personal appearance | Appearance personal neglect of |
| Neglect of personal appearance | Neglect of person appearance |
| Neglect of personal appearance | Neglect of personal appearance |
| Neglect of personal appearance | Personal appearance neglect of |

| Preferred Term | Lowest Level Term |
|---|---|
| Depression and Suicide/Self-Injury: Depression (SM | IQ) (Exclude Suicide/Self-Injury) |
| Poor quality sleep | Light sleep |
| Poor quality sleep | Poor quality sleep |
| Poor quality sleep | Poor sleep |
| Poor quality sleep | Sleep restless |
| Poor quality sleep | Sleep unwell |
| Poor quality sleep | Wakefulness |
| Psychomotor hyperactivity | Activity motor exaggerated |
| Psychomotor hyperactivity | Behavior hyperactive |
| Psychomotor hyperactivity | Behaviour hyperactive |
| Psychomotor hyperactivity | Hyperactive |
| Psychomotor hyperactivity | Hyperactivity |
| Psychomotor hyperactivity | Increased activity. |
| Psychomotor hyperactivity | Irritable hyperkinesis |
| Psychomotor hyperactivity | Motor activity exaggerated |
| Psychomotor hyperactivity | Muscular hyperactivity |
| Psychomotor hyperactivity | Overactive |
| Psychomotor hyperactivity | Overactivity |
| Psychomotor hyperactivity | Psychomotor agitation |
| Psychomotor hyperactivity | Psychomotor excitability |
| Psychomotor hyperactivity | Psychomotor hyperactivity |
| Psychomotor retardation | Psychomotor retardation |
| Psychosocial support | Psychosocial counseling |
| Psychosocial support | Psychosocial support |
| Psychotherapy | Art therapy |
| Psychotherapy | Cognitive psychotherapy |
| Psychotherapy | Couples psychotherapy |
| Psychotherapy | Family psychotherapy |
| Psychotherapy | Group psychotherapy |
| Psychotherapy | Hippotherapy |
| Psychotherapy | Interpersonal psychotherapy |
| Psychotherapy | Play therapy |
| Psychotherapy | Psychotherapy |
| Psychotherapy | Supportive psychotherapy |

| Preferred Term | Lowest Level Term |
|---|---|
| Depression and Suicide/Self-Injury: Depression (SMQ) | (Exclude Suicide/Self-Injury) |
| Self esteem decreased | Self esteem decreased |
| Substance-induced mood disorder | Stimulant-induced mood disorder |
| Substance-induced mood disorder | Substance-induced mood disorder |
| Tearfulness | Tearfulness |
| Terminal insomnia | Awakening early |
| Terminal insomnia | Early morning awakening |
| Terminal insomnia | Terminal insomnia |

| Preferred Term | Lowest Level Term |
|---|---|
| Depression and Suicide/Self-Injury: Suicide/Self-Injury | y (SMQ) |
| Columbia suicide severity rating scale abnormal | Columbia suicide severity rating scale abnormal |
| Completed suicide | Accomplished suicide |
| Completed suicide | Completed suicide |
| Completed suicide | Suicide |
| Completed suicide | Stricide (accomplished) |
| Depression suicidal | Depression suicidal |
| Depression suicidal Depression suicidal Intentional overdose | Suicidal depression |
| Intentional overdose | Deliberate overdose |
| Intentional overdose | Drug overdose deliberate self-inflicted |
| Intentional overdose | Intentional overdose |
| Intentional overdose | Multiple drug overdose intentional |
| Intentional overdose | Non-accidental overdose |
| Intentional overdose | Overdose deliberate self-inflicted |
| Intentional overdose | Overdose intentional |
| Intentional self-injury | Deliberate self-harm |
| Intentional self-injury | Deliberate self-injury |
| Intentional self-injury | Intentional self-injury |
| Intentional self-injury | Parasuicide |
| Intentional self-injury | Repeated parasuicide |
| Intentional self-injury | Self inflicted laceration |
| Intentional self-injury | Self mutilation |

| Preferred Term | Lowest Level Term |
|---|---|
| Depression and Suicide/Self-Injury: Suicide/Self-Injury | (SMQ) |
| Attempted suicide | Deliberate poisoning |
| Attempted suicide | Poisoning deliberate |
| Poisoning deliberate | Poisoning deliberate |
| Poisoning deliberate | Poisoning deliberate self-inflicted |
| Self injurious behaviour | Self injurious behavior |
| Self injurious behaviour | Self injurious behavior without suicidal intent |
| Self injurious behaviour | Self injurious behaviour |
| Self injurious behaviour | Self injurious behaviour without suicidal intent |
| Self-injurious ideation | Self-injurious ideation |
| Self-injurious ideation | Thoughts of self harm |
| Suicidal behaviour | Preparatory actions toward imminent suicidal behavior |
| Suicidal behaviour | Preparatory actions toward imminent suicidal behaviour |
| Suicidal behaviour | Suicidal behavior |
| Suicidal behaviour | Suicidal behaviour |
| Suicidal behaviour | Suicide gesture |
| Suicidal ideation | Active suicidal ideation |
| Suicidal ideation | Death wishes |
| Suicidal ideation | Life weariness |
| Suicidal ideation | Passive suicidal ideation |
| Suicidal ideation | Suicidal ideation |
| Suicidal ideation | Suicidal intention |
| Suicidal ideation Suicidal ideation | Suicidal plans |
| Suicidal ideation | Suicidal tendency |
| Suicide attempt | Attempted suicide |
| Suicide attempt | Suicide attempt |
| Suicide attempt | Suicide attempt other than overdose |
| Suicide attempt | Unsuccessful suicide |